### Cover page

# Psilocybin-assisted Group Therapy for Demoralization in Long-term AIDS Survivors

NCT02950467

**Protocol and SAP** 

17 April 2018

## PSILOCYBIN-ASSISTED GROUP THERAPY FOR DEMORALIZATION IN LONG-TERM AIDS SURVIVORS

Protocol Number: CHR#15-17825 ClinicalTrials.gov: NCT02950467

**IND Number:** 133326

Research Advisory Panel of California: PR#1705H

**DEA:** RW0519857

**Study Drug:** Psilocybin (4-phosphoryloxy-N,N-dimethyltryptamine) **Study Psychotherapy:** Supportive-Expressive Group Therapy

Version Number: 1.3 Version Date: 03 April 2018

#### Principal Investigator (Sponsor-Investigator)

Josh Woolley, MD, PhD University of California San Francisco 401 Parnassus Ave San Francisco, CA 94143

Telephone: 415-221-4810x24117

Fax: 415-379-5667

E-mail: josh.woolley@ucsf.edu

### **Co-Investigators**

Brian Anderson, MD, MSc James Dilley, MD Christopher Stauffer, MD

### **Statistician**

Matthew Boden, PhD

### **Clinical Research Coordinator**

Brian Anderson, MD, MSc University of California San Francisco 401 Parnassus Ave, Rm 263San Francisco, CA 94143 brian.anderson@ucsf.edu Telephone: 415-476-7432

Fax: 415-502-6361

#### **Proprietary and Confidential**

The information in this document is considered privileged and confidential, and may not be disclosed to others except to the extent necessary to obtain Institutional Review Board approval and informed consent, or as required by Federal and State laws. Persons to whom this information is disclosed should be informed that this information is privileged and confidential and that it should not be further disclosed.

### **Abstract**

| Title | Psilocybin-Assisted Group Therapy for Demoralization in Long-term AIDS Survivors |
|---|---|
| Patient population | Gay-identified HIV-positive men ≥50 years old who were diagnosed with HIV prior to 1996. |
| Rationale for Study | Long-term AIDS Survivors (LTAS) are people living with HIV (PLH) who were diagnosed prior to the advent of combined antiretroviral therapy (ART) and, compared to their HIV seronegative peers, suffer higher rates of depression, anxiety, trauma exposure, substance use and risky sexual behaviors [1-6]. Prior to ART, people living with HIV were "end-of-life patients," then with advent of ART they became "chronically ill," and now many of them are re-approaching end-of-life status as their bodies age at an accelerated rate due to HIV infection, HIV therapies, HIV-associated non-AIDS conditions, or all of the above [7]. By 2014, 9,202 HIV-positive individuals living in San Francisco were older than 50 years old (58% of the city's HIV-positive population) [8]. Like "cancer survivors," AIDS survivors experience increased rates of psychological distress even long after their disease is controlled [9, 10]. LTAS are an emerging population whose mental health needs are under recognized and undertreated. |
| | Existential distress is a form of psychological suffering precipitated by the acute awareness of one's mortality [11]. Demoralization is one type of existential distress [12], and it is characterized by a sense of hopelessness, helplessness and a loss of meaning in life [13]. Demoralization is a well-characterized clinical syndrome that captures the form of psychological distress suffered by many LTAS [1, 14]. Demoralization is also a clinical construct well-suited for investigation as a hypothesized therapeutic benefit of psilocybin-assisted psychotherapy in a population with chronic existential distress, like LTAS. Because it is experienced as a loss of meaning, demoralization should theoretically be treatable with interventions that enhance meaning-making [15]. An investigational pharmacotherapy that is thought to potently enhance meaning-making is psilocybin [16, 17]. Recent trials of individual psilocybin-assisted psychotherapy for anxiety and depression in cancer patients have shown this intervention to be safe [18-20], and have found significant improvements in anxiety and depression lasting months after a single treatment [19, 20]. Such impressive results are thought to be mediated by two mechanisms: 1) Having a complete "mystical-type" experience under the influence of psilocybin [21], and 2) Subsequent enhanced social support in the weeks following the mystical experience [22]. It remains unknown how these impressive results may translate into other palliative care populations. |
| | Since the beginning of the HIV/AIDS epidemic, many psychotherapies for people living with HIV have been preferentially delivered as groups because of enhanced cost-effectiveness and the group format's unique clinical benefits with respect to the enhancement of social support in a population suffering high rates of isolation and loneliness [23]. This study will use the same standard psilocybin administration safety guidelines |

| Rationale for Study (continued) | as prior trials [24], but the psychotherapy sessions will employ a modified form of Supportive-Expressive Group Therapy (SEGT) [25]. SEGT is a widely used, manualized, evidence-based group intervention for existential distress in patients with life-threatening disease [26]. The current study will be the first modern study of psilocybin-assisted group psychotherapy. In the current study, the group psychotherapy format functions as a standardized context in which patients' experiences of social support can be objectively observed pre- and post-psilocybin. This is helpful because while prior trials of psilocybin-assisted psychotherapy evaluated clinical outcomes, they did not make use of validated measures of psychotherapeutic process. By administering psilocybin as an adjunct to SEGT, we will be able to explore quantitatively and qualitatively not only the intrapersonal, but also the interpersonal, therapeutic mechanisms catalyzed by psilocybin in LTAS suffering from demoralization. |
|---|---|
| Primary<br>Objective | To demonstrate the safety and feasibility of Psilocybin-Assisted Supportive-Expressive Group Therapy (PA-SEGT) for demoralization in LTAS. |
| Exploratory<br>Objectives | To explore the preliminary efficacy of PA-SEGT for improving demoralization, complicated grief, depression, anxiety, quality of life, functional social support, post-traumatic growth, openness to experience, mindfulness, social connection, nature relatedness and ART medication adherence in LTAS. |
| | To explore quantitatively and qualitatively the mechanisms through which PA-SEGT addresses existential distress in LTAS. |
| Study Design | Open-label mixed-methods pilot study of individual oral psilocybin drug sessions (with escalating dose) combined with an evidence-based, manualized brief group psychotherapy. |
| Number of patients | 36 (maximum, with a minimum of 8) |
| Duration of<br>Therapy | 8 weeks after the initiation of the intervention. |
| Duration of Follow up | 3 months after completion of the intervention. |
| Duration of study | 2 years from the time the study opens to accrual. |
| Study Therapy | Psilocybin (4-phosphoryloxy-N,N-dimethyltryptamine) will be administered once at a moderate-to-high dose of 0.3mg/kg (or 0.36mg/kg) po during an individual medication visit to be held after 4 group therapy visits have been completed. Patients will undergo a total of 10 group psychotherapy sessions. |

Phase I – Study drug(s)


| Safety | Adverse events |
|---|---|
| Assessments | Vital signs |
| | Adverse Event Medication Session Form |
| | Columbia Suicide Severity Rating Scale Community Observer Rating Form |
| | Community Observer Rating Form |
| Feasibility | Rate of Patient Recruitment |
| Assessments | Rate of Patient Retention (Sessions Attended and Follow-ups Completed) |
| | Client Satisfaction Scale |
| | Individual Patient and Important Other/Caregiver Interviews |
| | Supportive-Expressive Group Therapy Topic Grid |
| | Focus Groups with Patients and Important Others/Caregivers |
| Primary<br>Outcomes | Demoralization Scale-II |
| Outcomes | Inventory of Complicated Grief |
| Secondary | Antiretroviral Medication Adherence Scale |
| Outcomes | Alcohol Use Disorders Identification Test |
| | Center for Epidemiologic Studies Depression Scale—Revised |
| | Challenging Experience Questionnaire |
| | Clinical Global Impressions Scale |
| | Credibility/Expectancy Questionnaire |
| | Duke/UNC Functional Social Support Questionnaire—5 |
| | Drug Use Disorders Identification Test |
| | Experiences in Close Relationships scale—Modified 16 |
| | Group Psychotherapy Intervention Rating Scale |
| | Group Questionnaire |
| | HIV and Abuse Related Shame Inventory |
| | Individual Group Member Interpersonal Process Scale |
| | International Personality Item Pool—Openness to Experience-20 |
| | McGill Quality of Life Questionnaire—Revised-Short |
| | Multidimensional Assessment of Interoceptive Awareness—Revised |
| | Mystical Experience Questionnaire—30 |
| | Nature Relatedness Scale, Short Form |
| | Post-traumatic Growth Inventory—Short Form |
| | PTSD Checklist-5 |
| | Schedule of Attitudes towards Hastened Death |
| | Social Connectedness Scale-Revised |
| | Outlai Cullifecteulless Scale-Neviseu |

Phase I – Study drug(s)


State-Trait Anxiety Inventory

Qualitative analysis of therapy sessions, interviews & focus groups

## Unique Aspects of this Study

This trial will be the first clinical trial of psilocybin-assisted psychotherapy for LTAS. It will also be the first modern trial of psilocybin-assisted group psychotherapy. It will be the first study of psilocybin-assisted psychotherapy for existential distress that will employ an evidence-based psychotherapy in the non-drug therapy sessions. The study will provide the first safety data for the use of this intervention in LTAS. It will not only yield preliminary data on the potential efficacy of this novel intervention. but it will also be the first study to employ both validated quantitative measures and qualitative methods in the analysis of the psychotherapeutic processes germane to psilocybin-assisted psychotherapy. It will also be the first clinical trial of psilocybin-assisted psychotherapy to assess the impact of the intervention on quality of life in partners/caregivers of LTAS. In anticipation of larger, better powered trials, clinical outcomes from this Phase I study will be used to produce the first estimates of effect size of this novel treatment for demoralization in palliative care patients.

Phase I – Study drug(s) 

#### **Table of Contents**

| 4 | _ | | | | | | | | | |
|---|---|-----|----|---|---|---|---|-----|---|---|
| 1 | 0 | ) [ | ni | r | വ | n | ш | cti | n | n |

- 1.1 Background on Indication
- 1.2 Background on Psilocybin-assisted Psychotherapy
- 1.3 Rationale for the Proposed Study
- 1.4 Study Hypotheses
- 2 Objectives of the Study
- 2.1 Objectives
- 2.1.1 Primary Objective
- 2.1.2 Exploratory Objectives
- 2.2 Endpoints
- 2.2.1 Primary Endpoints
- 2.2.2 Exploratory Endpoints
- 3 Study Design
- 3.1 Characteristics
- 3.2 Number of Subjects
- 3.3 Eligibility Criteria
- 3.3.1 Inclusion Criteria
- 3.3.2 Exclusion Criteria
- 3.4 Duration of Therapy
- 3.5 Duration of Follow Up
- 3.6 Randomization Procedures
- 3.7 Study Timeline
- 3.7.1 Primary Completion
- 3.7.2 Study Completion
- 4 Study Drugs
- 4.1 Description, Supply and Storage of Investigational Drugs
- 4.1.1 Investigational Drug: Psilocybin
- 4.2 Drug Accountability
- 4.3 Drug Ordering
- 4.4 Packaging and Labeling of Study Drugs
- 5 Treatment Plan
- 5.1 Dosage and Administration
- 5.1.1 Other Modalities
- 5.2 Monitoring and Toxicity Management
- 6 Study Procedures and Observations
- 6.1 Study Site
- 6.2 Selection of Measures
- 6.3 Qualitative Analyses
- 6.4 Schedule of Procedures and Observations
- 6.4.1 Phone Screening
- 6.4.2 In-person Screening and Enrollment
- 6.4.3 Baseline Assessments
- 6.4.3.1 Baseline Subject Assessments
- 6.4.3.2 Baseline Caregiver/Important others Assessments
- 6.4.4 Treatment Period
- 6.4.4.1 Week 1-4 Group Therapy Sessions

Phase I – Study drug(s) 

- 6.4.4.2 Weeks 5-6 Individual Drug Sessions
- 6.4.4.3 Weeks 7-10 Group Therapy Sessions
- 6.4.5 Endpoint Assessments
- 6.4.5.1 Endpoint (Week 10) Study Measures for Subject
- 6.4.5.2 Endpoint (Week 10) Study Measures for Caregivers/Important others
- 6.4.6 Post-treatment/Follow Up Assessments
- 6.4.6.1 Focus Group
- 6.4.6.2 3-Month Follow-up for Subject
- 6.4.6.3 3-Month Patients for Caregivers/Important others
- 6.4.6.4 3-Month Qualitative Interviews
- 6.5 Discontinuation of Therapy
- 6.6 Dietary Restrictions
- 6.7 Prohibited Medications
- 6.8 Study Clinicians
- 7 Reporting and Documentation of Results
- 7.1 Evaluation of Safety and Feasibility
- 7.2 Evaluation of Efficacy
- 7.3 Definitions of Adverse Events
- 7.3.1 Adverse Event
- 7.3.2 Adverse reaction
- 7.3.2.1 Suspected
- 7.3.2.2 Unexpected
- 7.3.2.3 Serious
- 7.3.2.4 Life-threatening
- 7.4 Recording of an Adverse Event
- 7.5 Follow-up of Adverse Events
- 7.6 Adverse Events Monitoring
- 7.7 Expedited Reporting
- 8 Statistical Considerations and Evaluation of Results
- 8.1 Study Design
- 8.1.1 Randomization
- 8.1.2 Stratification Factors
- 8.2 Determination of Sample Size and Accrual Rate
- 8.2.1 Sample Size and Power Estimate
- 8.2.2 Replacement Policy
- 8.2.3 Accrual estimates
- 8.3 Interim Analyses and Stopping Rules
- 8.4 Analyses Plans
- 8.4.1 Analysis Population
- 8.5 Primary Analysis
- 8.5.1 Exploratory Analyses
- 8.6 Study Results
- 9 Study Management
- 9.1 Pre-study Documentation
- 9.2 Institutional Review Board Approval
- 9.3 Informed Consent
- 9.4 Changes in the Protocol
- 9.5 Handling and Documentation of Clinical Supplies
- 9.6 Case Report Forms (CRFs)
- 9.7 Oversight and Monitoring Plan
- 9.8 Record Keeping and Record Retention

Phase I – Study drug(s) 

#### **Abbreviations**

AGPA American Group Psychotherapy Association

AHP Alliance Health Project

AIDS Acquired Immune Deficiency Syndrome

Albumin Alb

AlkPhos Alkaline phosphatase
Alt Alanine aminotransferase

AMAS Antiretroviral Medication Adherence Scale

AMAS ART Medication Adherence Scale

ANOVA Analysis of Variance
ART Antriretroviral Therapy
Ast Aspartate aminotransferase

AUDIT Alcohol Use Disorders Identification Test

BUN Blood Urine Nitrogen CBC Complete Blood Count

ChEQ Challenging Experience Questionnaire CrEQ Credibility/Expectancy Questionnaire

CESD-R Centers for Epidemiologic Studies Depression Scale—Revised

CHR Committee on Human Research
CMP Comprehensive Metabolic Panel
CORF Community Observer Rating Form

Cr Creatinine

CSS Client Satisfaction Scale

C-SSRS Columbia Suicide Severity Rating Scale CTC Concomitant Therapeutics Checklist

DEA Drug Enforcement Agency
DS-II Demoralization Scale—II
DSM Data and Safety Monitor

DUDIT Drug Use Disorders Identification Test

DUFSS-5 Duke UNC Functional Social Support Questionnaire-5

ECG Electrocardiogram

ECR-M16 Experiences in Close Relationships scale—Modified 16

ES Effect Size

FDA Food and Drug Administration

FT4 Free thyroxine

Gluc Glucose

GPIRS Group Psychotherapy Intervention Rating Scale

GQ Group Questionnaire

HAART Highly Active Antiretroviral Therapy

HANA HIV-Associated Non-AIDS

HARSI HIV and Abuse Related Shame Inventory

Hct Hematocrit Hgb Hemoglobin

HIM Hill Interaction Matrix

HIPPA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus ICC Intraclass Correlation Coefficient

ICF Informed Consent Form

ICG Inventory of Complicated Grief IND Investigational New Drug IOS Inclusion of Other in the Self

IPA Interpretive Phenomenological Analysis

IPIP-OE-20 International Personality Item Pool—Openness to Experience-20

LPPI Langley Porter Psychiatric Institute
LSD Lysergic acid diethylamide-25

Version date: 03 April 2018 Protocol CHR#15-17825

LTAS Long-term AIDS Survivor

MAIA Multidimensional Assessment of Interoceptive Awareness

MAOI Monoamine Oxidase Inhibitors

MEQ-30 Mystical Experience Questionnaire—30

MOCA Montreal Cognitive Assessment

MQoL-RS McGill Quality of Life Questionnaire—Revised-Short

NR Nature Relatedness Scale, Short Form NEO-PI-R Revised NEO Personality Inventory

OPLH Older People Living with HIV

PA-SEGT Psilocybin-assisted Supportive-Expressive Group Therapy

PCL-5 PTSD Checklist

PEQ-S Persisting Effects Questionnaire—Spirituality

PLH People Living with HIV

Plt Platelet

PPSv2 Palliative Performance Scale version 2

PTG Post-Traumatic Growth

PTGI-SF Post-Traumatic Growth Inventory—Short Form

PTSD Post-Traumatic Stress Disorder

QoLLTI-Fv2 Quality of Life in Life-Threatening Illness—Family Carer Version 2

SAHD Schedule of Attitudes towards Hastened Death

SCID-5-PD Structured Clinical Interview for DSM-5 Personality Disorders

SCID-5 Structured Clinical Interview for DSM-5 SCS-R Social Connectedness Scale-Revised SEGT Supportive-Expressive Group Therapy

SEGT-TG Supportive-Expressive Group Therapy Topic Grid SNRI Serotonin-Norepinephrine Reuptake Inhibitors

SSRI Serotonin Reuptake Inhibitors STAI State-Trait Anxiety Inventory

Tbili Total bilirubin

TCA Tricyclic Antidepressants

TProt Total protein

TSH Thyroid Stimulating Hormone

WBC White Blood Cell

Phase I – Study drug(s)


#### 1 Introduction

We propose to conduct a clinical trial of psilocybin-assisted psychotherapy for demoralization in Long-term AIDS Survivors (LTAS). This will be the first trial of psilocybin-assisted psychotherapy specifically for people living with HIV (PLH) and it will be the first modern trial of psilocybin-assisted *group* psychotherapy for any indication. The study will consist of three groups of six gay-identified HIV-seropositive men ≥50 years of age who were diagnosed with HIV prior to 1996 and who have moderate-tosevere demoralization [27] [13]. Each subject will undergo 8 weeks of a modified form of Supportive-Expressive Group Therapy [25] and one individual psilocybin treatment session [24] half-way through the intervention. Quantitative and qualitative measures of psychotherapeutic process will be used to explore the mechanisms by which this novel therapy seems to work, particularly on the interpersonal level. Quantitative and qualitative measures will assess changes in quality of life of the partners/caregivers of subjects undergoing the intervention. This study will contribute to the available data on the safety, feasibility and efficacy of psilocybin-assisted psychotherapy for existential distress in palliative care patients, and importantly will provide the first of such data on a palliative care population other than cancer patients [28].

Fig. 1 INTERVENTION TIMELINE



### 1.1 Background on Indication

Existential Distress and Demoralization

Existential distress is a form of psychological suffering that occurs when one is confronted with one's own mortality [11]. Demoralization is a form of existential distress that is prevalent in the palliative care setting and is characterized by hopelessness and helplessness due to a loss of purpose and meaning in life [12, 13]. Demoralization is associated with, but distinct from, depression, anxiety, isolation, and the desire for hastened death [29]. In palliative care patients, demoralization has been shown to be more strongly associated with suicidal ideation than depression is [30]. In modern palliative care, the current standard is to address existential and spiritual issues in patients and their family members [31, 32]. Following the lead of innovators like Frankl [33] and Yalom [34], investigators have over the last two decades devised a number of existential psychotherapies [35-40] with varying impact on depression, anxiety and quality of life

Phase I – Study drug(s) 

Version date: 03 April 2018

[26, 41]. Arguably, what these therapies have in common is what Cassel [42] long ago prescribed for the relief of suffering—*transcendence*—an experience that is difficult to define medically and a challenge to provide consistently in clinical settings. Palliative care stands to benefit greatly from a time-limited intervention that enhances patients' capacity to forge meaning, to transcend suffering, and to overcome social isolation and the fear of the unknown in a safe, immediate and reliable manner. This need is pronounced among LTAS.

#### **AIDS Survivors**

By 2004, there had been an estimated 929,985 cases of AIDS in the US, and 524,060 of them had died [43]. With the advent of combined antiretroviral therapy (ART) in 1996, HIV seropositive individuals began to accomplish what once was thought to be impossible—living into old age. Because of the decreased lifespan and the apparently accelerated aging experienced by PLH, "older" in HIV is defined as ≥50 years of age [44]. Many LTAS are therefore also considered older people living with HIV (OPLH). Despite recent gains in mortality, many of today's LTAS are still grappling with having been, at one point, an "end-of-life" patient. Beyond being confronted by their own mortality at the time of diagnosis, LTAS frequently bore witness to the deaths of friends and loved-ones, and often served as informal caregivers to those dying of AIDS [45]. AIDS-related bereavement is associated with demoralization, depression, and problematic substance use [46]. Survivor's guilt is common among LTAS, as is loneliness [47]. Isolation and loneliness are highly prevalent among LTAS not only because the gay community was decimated by AIDS in the 1980s and '90s, but also because many OPLH often lack traditional family support structures due to several possible causes that include protective withdrawal from one's biological family, having been disowned by family or friends due to stigma, or not having children [1, 47]. Because of reduced social support networks, and therefore a relative lack of access to informal caregivers, OPLH are in general expected to be especially reliant on community-based services as they age [1].

#### Multimorbidities

Compared to HIV seronegative demographically- and behaviorally-matched peers, OPLH are at increased risk of multimorbidities known as HIV-associated non-AIDS (HANA) conditions. such as cardiac disease, with PLH having a 50% increased risk of acute myocardial infarction compared to HIV seronegative matched controls [48]. PLH are also at higher risk of some HANA malignancies, having three times the cumulative incidence of liver cancer and thirty times the cumulative incidence of anal cancer [49]. PLH are also at increased risk of serious bone, liver and kidney disease [44, 50]. As the health of OPLH declines, HANA and other conditions can serve as continual reminders of one's mortality. OPLH also suffer from high rates of mental health conditions such as depression (prevalence up to 50%), suicidal ideation, and anxiety (prevalence up to 20%) [1, 2]. AIDS patients have been found to have an increased desire for hastened death [51]. Among PLH (of all ages) PTSD has a prevalence that ranges 10-74% [3, 52]. Like PLH of other ages, OPLH have higher rates of substance use [4, 5, 53] and risky sexual behaviors [6] than the general population and these behaviors are associated with ART nonadherence and therefore disease progression and secondary HIV transmission [54]. The incidence of HIV in US adults over 50 years of age saw no improvement from 2010-2014 [55]. Comorbid depression, anxiety and PTSD are also associated with ART non-adherence in PLH [56-59]. Depression treatment has been shown to increase ART adherence in PLH [60], and possibly to decrease secondary transmission of HIV [61]. Data specific to OPLH and behavioral interventions that increase ART adherence, however, is limited to few studies that are wanting in methodological rigor [62].

#### Older People Living with HIV

The CDC projected that people over the age of 50 years would constitute the majority of the HIV-positive population in the US by 2015 [63]. OPLH became the majority of the HIV-positive population in San Francisco in 2012, and their proportion of the population continues to rise [8].

Phase I – Study drug(s) 

It is estimated that over 70% of the US HIV seropositive population will be ≥50 by 2020 [64]. The NIH Office of AIDS Research Working Group on HIV and Aging has highlighted as priority research areas, among others: Research on mental health in older adults with HIV and possible interventions; Research on substance use in older adults with HIV; Research on social networks and care giving of older adults with HIV [1]. The HIV community has responded to the demographic change by forming peer support groups and holding town halls on the issue across the country [65]. Organizational initiatives have sprung up around the issue, including patient advocacy groups like the Medius Institute and Let's Kick AIDS Survivor Syndrome (www.letskickass.org), with "AIDS Survivor Syndrome" being a patient-promoted syndrome characterized by traumatic exposure, complicated grief, depression, self-destructive behavior and hopelessness. Also, many local government and non-profit efforts have emerged over the last half decade, including the AIDS Community Research Institute of America's Center on HIV and Aging, the 50-Plus Program at San Francisco AIDS Foundation, and the San Francisco County Workgroup on HIV and Aging. Finally, the popular press has recently directed attention to the issue [66-68], and in 2016 the San Francisco Chronicle even made a feature-length documentary on the struggles of older HIV-positive gay men in San Francisco [69].

#### Treatment Needs

Much of the recent literature on the mental health treatment needs of OPLH has focused on depression [7]. Despite the well-established relationship between depression, grief and demoralization in PLH [46], grief and demoralization have been less frequently studied since the advent of combined ART. Preliminary analysis of outcomes from support groups for OPLH at UCSF's Alliance Health Project (AHP) indicates that depression and anxiety symptoms improve from participating in these groups, but trauma symptoms, particularly related to traumatic losses, tend to persist [70]. These AHP findings are supported by the literature that shows that coping/support groups for OPLH can improve depressive symptoms [71]. This is also supported by anecdotal evidence from the Director of the San Francisco AIDS Foundation's 50-Plus program, who reports that members of this community need more access to treatments for psychological trauma [65]. Current literature suggests that PLH have difficulty finding therapies that adequately address traumatic loss and grief [72]. More specifically, the Director of the San Francisco AIDS Foundation's 50-Plus program has stated "We need a treatment tailored to our community's needs; not just recycled therapies for other people," which again is supported by the literature which suggests that PLH respond better to therapies specifically targeted to grief and psychiatric distress (done in a group) than generic individual psychotherapy [73]. Whereas coping groups for bereavement in PLH have shown brief but unsustained improvements in grief, they have not proven to benefit general psychological distress or functioning [43]. Another recent study did demonstrate short-term reductions in traumatic stress from a coping group intervention in PLH, but no data are available on the durability of these benefits [74].

#### Group Therapy, Social Support, and Post-Traumatic Growth

Spiegel and Yalom's Supportive Expressive Group Therapy (SEGT) [34, 75] was originally designed as an intervention for advanced cancer patients, has since been modified to be used with a variety of palliative care patients, and has a robust evidence base for its efficacy [41]. SEGT emphasizes social support and increasing communication with caregivers. It also focuses on processing affect in the 'here and now' and 'detoxifying death and dying'; it includes exposure to a therapeutic altered state of consciousness (self-hypnosis); and it encourages emotional expression and openness [25]. Manuals exist for traditional (1 year) [75] and brief (12-week) [76] SEGT, and SEGT has been shown to be teachable [77]. SEGT has also already been modified for and used with success in patients with advanced HIV [78]. A recent study of tele-SEGT for depressed OPLH found that therapeutic alliance did not predict clinical response, but group cohesion and perceived member similarity did [79]. Social support in PLH is related to improved mood, well-being and medication adherence [44]. Enhanced social support in PLH is also associated with enhanced post-traumatic growth (PTG) [80]. Whereas much of the literature on

Phase I – Study drug(s) 

the mental health of PLH focuses on coping, the concept of PTG goes beyond coping with the problems associated with living with HIV and includes improvement in one's mental health. PTG comprises an increased appreciation for life, enhanced self-efficacy and ability to forge intimate relationships, and the increased expression of emotions and hope for the future [80]. PTG is associated with fewer depressive symptoms in PLH [81]. Currently, however, there is a dearth of literature specifically on PTG and HIV [3, 82], especially on interventions that enhance it. Of particular relevance to our study, PTG is associated with a heightened interest in spirituality [80].

#### Psychoneuroimmunology in HIV

It seems that HIV remains a rich field of investigation of the mind-body connection, and perhaps especially among OPLH who may have greater mental and physical health needs compared to younger PLH. Earlier literature on psychoneuroimmunology and HIV regularly found associations between depression, traumatic exposure and disease progression and mortality in PLH, both before and soon after the advent of highly active antiretroviral therapy (HAART) [83, 84]. It is unclear whether such associations remain with the improved ART regimens available today. Nevertheless, recent data have shown that spiritual coping in PLH is associated with increased survival [85]. And after controlling for ART use, depression, hopelessness, and avoidant coping have predicted the progression of viral load and CD4 count longitudinally [86]. Recent data from the NIH indicate that PTSD is associated with differential immune activation in PLH, even in those who are virally suppressed [52]. While spirituality and religiosity have been positively associated with enhanced mental health in PLH, the personality traits of conscientiousness, openness and agreeableness (measured with the NEO-PI-R) are more strongly positively associated with mental health in this population [87]. Openness has also been inversely associated with disease progression over 4 years [88]. Finally, in PLH dispositional mindfulness has been inversely related to depression, stress appraisal and negative affect, while it is positively associated with positive affect [89].

### 1.2 Background on Psilocybin-assisted Psychotherapy

Psilocybin is a natural product found in many species of psychoactive fungi around the world [90]. Modern scientific research with psilocybin began when the chemist Albert Hoffman first isolated psilocybin from *Psilocybe mexicana* mushrooms in 1957 [91]. Psilocybin (4-phosphoryloxy-N,N-dimethyltryptamine) is the prodrug of psilocin (4-hydroxy-N,N-dimethyltryptamine), an indoleamine that acts as an agonist of serotonin 5HT 1A, 2A and 2C receptors [92]. In humans, psilocybin is rapidly metabolized to psilocin after oral ingestion; psilocin has no known P450 interactions and is instead glucoronidated and renally excreted [91, 93, 94]. Relative to other psychedelics (e.g., lysergic acid diethylamide-25, a.k.a. LSD), psilocybin has a simpler neurotransmitter receptor profile (it is known to act only at serotonin receptors) and a shorter duration of acute effects (4-5 hours) [91, 95]. Psilocybin is one of the "classic hallucinogens" (a.k.a. "classic psychedelics") that were investigated in the mid-20<sup>th</sup> century for their potential as pharmacologic adjuncts to psychotherapy. By the mid-1960s, over 1,000 clinical reports were published on the experiences of over 40,000 treatment sessions in which psychedelics had been legally administered to patients in clinical settings [96] such as at Harvard [97], UCLA [98], and UCSF [99].

This early research suggested that one of the most promising indications for psychedelic-assisted psychotherapy was the treatment of existential distress in patients with advanced disease, particularly cancer. This was first reported by Kast, an internist who administered LSD (without psychotherapy) to terminally-ill patients as an experimental analgesic. He found that a single dose of LSD decreased physical discomfort and improved mood, and that these effects lasted for about 10 days [100]. More systematic work later occurred at Spring Grove Hospital near Baltimore, Maryland where a team developed a protocol for psychedelic-assisted psychotherapy for the terminally ill. Their protocol included several non-drug preparatory

sessions designed to build trust and rapport between the participant and the therapists. Then, during the drug session itself, the therapists (usually a team of two) would sit beside the patient and mostly provided non-directive verbal reassurance. Afterward, several non-drug psychotherapy follow-up sessions took place over the next few weeks to psychologically "integrate" the drug experience into the patient's life. One legacy of this work is the safety protocol recently developed at Johns Hopkins [24] for psychedelic drug administration, which has been adapted for this proposed study.

In the 1970s, before rigorous and well-controlled trials of the Spring Grove protocol could be undertaken, clinical research with psychedelics in the US was abandoned due to increased regulatory requirements and an unfavorable political climate. Nevertheless, pharmacology and neuroscience studies continued, producing a clear understanding of psilocybin's effects on neurotransmitter receptors and human physiology [91, 92, 101]. Unlike many other Schedule I controlled substances, the "classic psychedelics" are physiologically safe over a wide range of doses and have a low potential risk of addiction [92, 102]. The published case series of mid-Century psychedelic-assisted psychotherapy reveal an overall low rate of adverse events when administered in controlled clinical settings [103]. (For more clinical safety data, see Section 4.1.1 below.) And while clinical research ceased in the US in the 1970s, psilocybin-assisted individual and group psychotherapy continued to be practiced legally in Germany and Switzerland into the 1990s [104].

Clinical research with psychedelics in the US reemerged in the 1990s when Strassman investigated the pharmacology of dimethyltryptamine in healthy volunteers [105]. He was followed by Griffiths et al who conducted a double-blinded RCT in which healthy volunteers were administered a single high dose of psilocybin (0.43mg/kg) vs active placebo (methylphenidate) and found that a significantly higher proportion of volunteers receiving psilocybin had "complete mystical experiences" [17]. Seventy-four percent of subjects rated the psilocybin experience as one of the five most spiritually significant experiences of their lives (compared to 8% of controls) [17]. Remarkably, subjects who received psilocybin also demonstrated significant increases in the personality trait of Openness on the NEO-Personality Inventory (e.g., aesthetic appreciation and sensitivity, imagination and fantasy, and tolerance of others' views and values) 12 months after drug administration. No other discrete clinical intervention has ever been shown to cause significant and enduring changes in an adult's personality structure [106].

The Griffiths et al. 2006 study was followed by Grob et al [18], who demonstrated in a doubleblind cross-over RCT the safety and feasibility of psilocybin-assisted psychotherapy in 12 advanced cancer patients with a DSM-IV anxiety diagnosis deemed to be secondary to their cancer diagnosis. This study utilized a single moderate dose of oral psilocybin (0.2mg/kg), and found improvements in anxiety and depression in the months following the intervention. The most recent data on psilocybin-assisted psychotherapy in existential distress in cancer patients come from two recently completed Phase II trials, whose results have not yet been published: Ross et al. conducted a double-blind cross-over RCT comparing an active placebo (niacin) to a single high dose of oral psilocybin (0.3mg/kg) in 29 cancer patients with moderate-to-severe anxiety and whose cancer was either active or in remission with a chance of recurrence. Their study found significantly greater reductions in anxiety and depression with psilocybin (versus placebo) lasting from hours after the drug session to up to 8 months later [19]. The second study, conducted by Griffiths et al, was a double-blind, cross-over RCT comparing a subthreshold dose (0.014) to a moderate-to-high dose (0.31) oral psilocybin in 51 cancer patients with depression and anxiety. They found reductions in anxiety and depression (both within-group and between groups) that were significant at 5 weeks post-treatment; the improvements in mood persisted at the 6 month follow-up time point [20].

Over the past 20 years psilocybin has shown to be safe and preliminarily effective in the treatment of not only existential distress in cancer patients [18-20], but also treatment-resistant

alcohol use disorder [107], treatment-resistant tobacco use disorder [108, 109], and obsessive-compulsive disorder [110].

#### 1.3 Rationale for the Proposed Study

Rationale for Psilocybin-Assisted Psychotherapy for Demoralization in LTAS Per Section 1.1. above, there is a large unmet need for the treatment of existential distress in LTAS. Compared to classic examples of acute existential distress in end-of-life patients (e.g., cancer patients or advanced AIDS patients), the existential distress of LTAS is a more chronic condition complicated by severe grief and traumatic exposure. Like "cancer survivors." AIDS survivors often experience increased rates of psychological distress long after their disease is controlled [9, 10]. While the existential distress of LTAS is multifaceted and complex, the wellcharacterized clinical syndrome of demoralization appears to capture the type of psychological distress suffered by many LTAS (6, 7). The concept of demoralization is predicated on the loss of one's meaning-making ability in the face of distress. Enhancing meaning-making to address existential distress and complicated grief is a strategy that has been embraced not only by palliative speciatlists [36] and thanatologists [15], but also by the HIV community itself [65]. In general, the mental health needs of LTAS —an emerging, medically and psychosocially complex, and stigmatized population—remain under-recognized and undertreated, but in particular it seems LTAS could benefit from a brief intervention that would enhance meaningmaking in order to better cope with, and transcend, years of loss and suffering.

Modern studies of psilocybin-assisted psychotherapy for cancer patients and cancer survivors with existential distress provide promising preliminary evidence of this intervention in treating demoralization in palliative care patients [18-20]. These clinical improvements are thought to be mediated by having a complete "mystical-type" experience [21], which leads to an enhanced sense of meaning in one's life [111], and an enhanced ability to engage with one's social supports [22]. Moreover, psilocybin may also help improve patients' relationships with love-ones who have already died: According to the most experienced clinician in the field of psilocybin-assisted psychotherapy, Dr. William Richards (who began treating palliative care patients with this method in the 1970s), psilocybin-assisted psychotherapy can be highly effective at treating protracted grief [112]—a rather difficult to treat symptom in LTAS (see above, Section 1.1 Treatment Needs).

LTAS – An Ideal Model for Studying Chronic Existential Distress in Palliative Care Patients
Clinical trials in palliative care are fraught with many methodological challenges, especially
subject recruitment given patients' lack of interest in spending their limited time in research
studies, or inability to comply with the physical demands of attending study visits and research
protocols [113]. Attrition rates of up to 50% are not uncommon among psychotherapy trials with
palliative care patients [77, 114, 115]. Recent trials of psilocybin-assisted psychotherapy for
existential distress in cancer patients have struggled with recruitment [28]. The current proposed
study of psilocybin-assisted psychotherapy in LTAS is unlikely to be hindered by these same
recruitment challenges because the form of existential distress to be examined, demoralization,
is thought to occur at high rates [65] among a largely ambulatory population that is known to
avidly volunteer for medical research [116] and is desperately in search of treatment options
[65]. Despite the fact that HIV is now considered a "chronic illness" and not an acutely lifethreatening condition for most patients, PLH potentially face their mortality on a daily basis when
they choose, or choose not, to adhere with their ART regimen, thus likely enhancing existential
distress chronically.

Rationale for using Psilocybin as a Psychotherapy Adjunct, and eschewing Psilocybin Monotherapy

This trial does not include a control arm of psilocybin without psychotherapy. When psilocybin and other psychedelics were investigated as pharmacologic adjuncts to psychotherapy in the 1950s and 60s, clinical experience led to the principle of "drug, set and setting," [117] which states that the clinical safety and outcomes of a psychedelic drug experience are highly influenced by the non-pharmacological variables of the patient's mental state prior to drug administration ("set") and their environment during the experience ("setting"). Unlike other modalities of drug-assisted psychotherapy (e.g., D-cycloserine-assisted cognitive behavioral therapy), in psychedelic-assisted psychotherapy, not only is the drug experience thought to deeply influence the content of the psychotherapy, but the content of the psychotherapy is likewise understood to intimately shape the drug experience itself. This consideration has led to the consensus that it is unethical for psychedelics to be administered to patients absent a supportive and therapeutic context. This context has typically been individual psychotherapy, but group therapy modalities have also been used. [96, 118]

#### Rationale for Group Therapy

Since the beginning of the HIV/AIDS epidemic, many psychotherapies for PLH have been preferentially delivered as groups because of enhanced cost-effectiveness and the group format's unique clinical benefits with respect to the enhancement of social support in a population suffering high rates of isolation and loneliness [23].

The theoretical basis of the original Spring Grove approach to treating existential distress in palliative care patients was that patients suffer extreme *isolation* because of their disease, and that psychedelic-assisted psychotherapy could help relieve this isolation by facilitating: 1) living meaningfully in the present moment, and 2) reaching out and authentically connecting with loved ones [22]. Various clinical benefits were reported from their uncontrolled experimental sessions, including improvements in mood and anxiety, and increased openness to communication with loved ones [119]. These older findings are consistent with more recent social psychology findings that psilocybin decreases the subjective feeling of social exclusion [120] and another classic psychedelic, LSD, enhances emotional empathy and prosocial behavior [121].

The Spring Grove team concluded that optimal clinical outcomes were dependent upon attaining a "psychedelic peak experience," which was conceived of as akin to William James' "conversion experience," [122] or Abraham Maslow's "peak experience," [123] —a transcendent state of unity, intense positive emotions, and ineffability that was experienced as deeply meaningful. [22] To describe this mental state, the current psilocybin literature has adopted the terminology of the "complete mystical experience," which is defined by standard criteria using a validated psychometric measure, the Mystical Experience Questionnaire—30 item [124]. Because the Spring Grove team believed that the "transcendental nature of the experience [could] neutralize a sense of alienation..." they sought to facilitate such experiences in order "to maximize patients' opportunities for living by lessening their sense of isolation and alienation. and in so doing, assist in their reaching out to those around them" [125]. One aspect of this model that has received little mention in the recent literature is that the original Spring Grove protocol included non-drug family therapy sessions conducted both before and after drug sessions [22]. The purpose of these sessions was to prepare the family to better help the patients integrate their psychedelic experience after the drug sessions, as well as to aid the family in their imminent grieving process.

Spontaneous feedback from several subjects in the recent NYU psilocybin-assisted psychotherapy trial for existential distress in cancer patients included the request to be introduced to the other study subjects [19], apparently to share, process and integrate their experiences in a setting of mutual aid and understanding. Subjects from recent MDMA-assisted psychotherapy trials for PTSD have also spontaneously made this request, leading the study


Version date: 03 April 2018

sponsors to create a web forum for the patients to be in touch with each other after completing the trials [126]. It appears to be helpful to patients treated with psychedelic-assisted psychotherapy to spend time with peers in their attempt to integrate the "peak" experiences, the phenomenology of which can be rather uncanny and perhaps difficult for psychedelic-naïve family or friends to comprehend [127].

Conducting non-drug psychotherapy sessions in groups may shed light on possible key mechanisms of psilocybin-assisted psychotherapy for existential distress. Whereas *therapeutic alliance* is thought to be the most important mediator of clinical outcomes in individual psychotherapy, *group cohesion* is widely recognized as the analogous mechanism in group psychotherapy [128, 129]. Examining the change of group cohesion pre- and post-psilocybin with validated self-report [130] and observer-rated instruments [131] will provide a novel and standardized means of observing how psilocybin drug sessions may affect the interpersonal functioning of distressed palliative care patients.

A significant limitation of group therapy clinical trials is that large sample sizes are required to demonstrate efficacy because of the likely interdependence of outcomes of members of the same group [132]. For this reason, qualitative (e.g. Interpretive Phenomenological Analysis) and/or sequential (e.g. the Hill Interaction Matrix) measures of psychotherapeutic *process* are often used to make inductive inferences about clinical change from group therapy over time [133]. Process is understood as the conglomeration of intrapersonal functions, interpersonal dynamics and group environment that leads to therapeutic change [134]. To improve the evidence base for group psychotherapy, the American Group Psychotherapy Association (AGPA) has developed clinical practice guidelines [135] and a standard set of measures and tools for creating and managing psychotherapy groups for clinical practice and research [136]. In developing the protocol for this proposed study, we have drawn not only from the literatures on psilocybin-assisted psychotherapy and palliative care, but also from these AGPA clinical and research guidelines, as well as on the consultation of local group psychotherapy experts [137].

#### Rationale for Dosing Regimen

Griffiths et al [138] have characterized the dose-response relationship of oral psilocybin in healthy volunteers. They found that when considering the odds of attaining a complete mystical experience versus having a temporary anxiety reaction during the drug experience (lasting on the order of minutes), the optimal dose likely falls between 0.29mg/kg and 0.43mg/kg [138]. This dose range has been successfully used in studies of psilocybin-assisted psychotherapy for existential distress in cancer patients [19, 20], severe alcohol use disorder [107] and tobacco use disorder [108]. The current study will employ a dose of 0.3mg/kg po in the first group, and if this is well tolerated will then escalate to 0.36mg/kg po in subsequent groups.

The dosing of the psychotherapy—8 weekly sessions—was chosen on the basis of comparison with similar group psychotherapies for existential distress in palliative care patients. The group psychotherapy with the best evidence-base for treating existential distress in palliative care patients, Meaning-Centered Group Psychotherapy, also employs 8 sessions [139]. The group psychotherapy with the best evidence-based for treating complicated grief has 16 weekly sessions [140]. Our protocol uses a modified course of Brief Supportive-Expressive Group Therapy, which was designed and tested as a 12-week course of treatment [76]. Empirical data suggest that group therapies lasting at least 12 sessions are shown to have greater correlations between group cohesion and clinical outcomes [129]. We hypothesize that psilocybin will catalyze group cohesion in a shorter period of time, thus making 12-16 weeks of group therapy unnecessary for detecting comparable results with regards to cohesion and clinical outcomes.

Rationale for Supportive-Expressive Group Therapy

Version date: 03 April 2018 Protocol CHR#15-17825

While prior trials of psilocybin-assisted psychotherapy for existential distress in palliative care patients have followed a standard drug administration safety protocol, they have not used manualized psychotherapies in the non-drug therapy sessions; our study will be the first to do this, which should enhance generalizability of the results. The format and content of SEGT are appropriately flexible for incorporating individual psilocybin sessions during the course of therapy, and including psychoeducation on psilocybin in the preparatory sessions. The focus of SEGT on expressing emotions and enhancing communication with caregivers is expected to be helpful in integrating psilocybin experiences [118]. Psilocybin has been shown to enhance access to positive emotional memories [141] and to increase the personality trait of openness [106], and this should support SEGT's aim of increasing awareness of one's emotions and openness to new experiences. Because the primary aim of this pilot trial is to assess safety and feasibility of this modality—and assessing efficacy is a secondary aim—no control group of traditional SEGT will be included in the study. For the rationale on why psilocybin monotherapy (without an adjunctive psychotherapy) will not be offered as control condition, see above.

### 1.4 Study Hypotheses

#### Primary

1. The study will recruit, consent and enroll at least 18 subjects (in 3 groups of 6 members) over 18 months; these subjects will complete all treatment and evaluation sessions and they will experience no treatment-emergent serious adverse events.

#### Secondary

- The difference in pre- and post-treatment mean scores of demoralization, complicated grief, depression, PTSD, shame, anxiety, quality of life, functional social support, posttraumatic growth, openness to experience, attachment security, mindfulness, global clinical impressions and ART medication adherence will trend toward significant improvement. These improvements will be sustained at 3-month follow-up.
- 2. The difference in pre- and post-psilocybin rates of change of group cohesion and group process will trend toward significant improvement.
- 3. Qualitative analyses of subject behavior and caregiver/important other reports will lead to greater understanding of the interpersonal mechanisms of action of psilocybin-assisted psychotherapy.

### 2 Objectives of the Study

#### 2.1 Objectives

#### 2.1.1 Primary Objective

 To demonstrate the safety and feasibility of Psilocybin-Assisted Supportive-Expressive Group Psychotherapy (PA-SEGT) for demoralization in long-term AIDS survivors (LTAS).

#### 2.1.2 Exploratory Objectives

- To explore the preliminary efficacy of PA-SEGT for improving demoralization, complicated grief, depression, PTSD, shame, anxiety, post-traumatic growth, quality of life, functional social support, openness to experience, attachment security, social connection, nature relatedness and ART medication adherence in LTAS.
- To explore quantitatively and qualitatively the mechanisms (e.g. group cohesion) through which PA-SEGT addresses demoralization and other mental health outcomes in LTAS.

### 2.2 Endpoints

#### 2.2.1 Primary Endpoints

- Safety will be defined based on the rate of adverse reactions (defined by the NIH Division of AIDS Table of Grading of Severity of Adult and Pediatric Adverse Events V2.0) (see Section 5 below). The safety of acute drug effects will be assessed by monitoring vital signs for tachycardia (HR>100bpm), bradycardia (HR<60bpm), hypertension (SBP>140mmHg or DBP>90mmHg) and hypotension (SBP<100mmHg or DBP<60mmHg). Drug-induced mental status changes will be assessed using the Adverse Event Medication Session Rating Form during drug sessions, pre and post measures with the Montreal Cognitive Assessment, and the Persisting Effects Questionnaire—Spirituality at study follow up. Suicidality will be assessed with the Columbia Suicide Severity Rating Scale. Follow-up safety data will be gathered for 3 months.</li>
- Feasibility will partially be assessed in terms of the rates of patient recruitment and
  retention. Feedback on acceptability will also be gathered from subjects and
  caregivers/important others using the Client Satisfaction Scale. Patients and caregivers
  will also be invited to provide feedback during a focus group and patients will be invited
  to participate in individual interviews after the intervention. A SEGT Topic Grid will be
  used to evaluate video recordings of group therapy sessions in order to assess therapist
  adherence to the PA-SEGT model.

### 2.2.2 Exploratory Endpoints

Preliminary efficacy will be assessed with the primary clinical outcome measures:

- Change in demoralization will be defined as the difference in pre-treatment, post-treatment, and 3-month follow-up scores of the Demoralization Scale-II.
- Change in complicated grief will be defined by the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of the Inventory of Complicated Grief.

Preliminary efficacy will also be explored with the following secondary endpoints (See Section 5 for details on individual measures):

- Change in ART medication adherence will be defined as the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of the ART Medication Adherence Scale.
- Change in depression will be defined by the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of the Center for Epidemiologic Studies Depression Scale—Revised. Change in subject quality of life will be defined by the difference in pre-treatment, post- treatment, and 3-month follow-up mean scores of the McGill Quality of Life Questionnaire—Revised.
- Change in desire for hastened death will be defined as the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of Schedule of Attitudes towards Hastened Death.
- Change in anxiety will be defined as the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of the State-Trait Anxiety Inventory.
- Change in social support will be defined as the difference in pre-treatment, posttreatment, and 3-month follow-up mean scores of the Duke/UNC Functional Social Support Questionnaire-5.
- Post-traumatic growth due to the intervention will be defined by post-treatment and 3month follow-up mean scores of Post-Traumatic Growth Inventory—Short Form.
- Change in PTSD symptoms will be defined as the difference in pre-treatment, post- treatment, and 3-month follow-up mean scores of the PTSD Checklist-5.
- Change in global clinical status will be defined as the difference in pre-treatment and post- treatment mean scores of the Clinical Global Impressions Scale completed by an clinical rater.
- Change in openness to experience will be defined as the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of the International Personality Item Pool—Openness to Experience-20 scale.
- Change in mindfulness will be defined as the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of subscales of the Multidimensional Assessment of Interoceptive Awareness.
- Change in social connectedness will be defined by the difference in pre-treatment, posttreatment, and 3-month follow-up mean scores of the Social Connectedness Scale— Revised.
- Change in Nature Relatedness will be defined by the difference in pre-treatment, post-treatment, and 3-month follow-up mean scores of the Nature Relatedness Scale, Short Form Version.
- Change in alcohol and drug use will be defined by different in the baseline and 3-month follow-up AUDIT and DUDIT scores

Psychotherapeutic process and mechanisms will be explored with the following endpoints:

- Change in group cohesion will be defined as the difference in rate of Group Questionnaire score change pre- and post-psilocybin.
- Change in group process will be assessed as the difference in rate of progression of

Phase I – Study drug(s) 

the Hill Interaction Matrix score pre- and post-psilocybin.

- Change in group process will be assessed as the change in the Individual Group Member Interpersonal Process Scale over time.
- Expectancy effects will be estimated based on the pre-psilocybin total score of the Credibility/Expectancy Questionnaire.
- Subjective experience of a psilocybin treatment session will be evaluated with the Mystical Experience Questionnaire—30 and the Challenging Experience Questionnaire.
- Change in attachment security will be defined as the difference in pre-treatment, posttreatment, and 3-month follow-up mean scores of the Experiences in Close Relationships scale—Modified 16.
- Qualitative analysis of therapy session video footage, semi-structured patient interviews, focus groups and process notes written by study staff.
- Change in inclusion of other in self will be defined by the difference in pretreatment, post-treatment, and 3-month follow-up results of the Inclusion of Other in Self measure.

Phase I – Study drug(s) 

### 3 Study Design

Version date: 03 April 2018

#### 3.1 Characteristics

This is a Phase I open-label pilot mixed-methods study of the safety and feasibility of an 8-week group psychotherapy intervention that includes one individual drug session with oral synthetic psilocybin. This intervention is designed to treat demoralization in LTAS. Groups of 6 subjects will be run in sequence. Safety data will be gathered before, during, immediately after, and for 3 months after the intervention. Subjects will complete self-report measures and semi-structured interviews related to acceptability and subjective experience. Exploratory analyses will be conducted of clinical outcomes. Exploratory analyses will also include quantitative and qualitative assessments of psychotherapeutic process mechanisms.

### 3.2 Number of Subjects

We estimate that a total of 60 patients will be screened in-person for the study. We estimate that at least 18 patients will need to be enrolled given the high rate of drop outs seen in group psychotherapy studies in this population [114]. Patients who have been assigned to a group will be replaced only if they drop out prior to the first group therapy session (this avoids the possible symbolic message that if a subject were to die, that he would be easily replaced in the group). We aim for, at minimum, 8 subjects (two groups of at least 4 subjects each) will complete the study; at maximum, 36 subjects (six groups of six subjects each) will complete the study. (See Section 8.2.1 Sample Size and Power Estimate.)

### 3.3 Eligibility Criteria

Patients must have baseline evaluations performed prior to the first group therapy session and must satisfy all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified.

#### 3.3.1 Inclusion Criteria

- 1. Gay-identified men ≥50 years old who are able to understand a written informed consent document and who are willing to sign it.
- 2. Laboratory confirmed HIV seropositive status; and diagnosed prior to 1996.
- 3. Moderate-to-severe demoralization, determined by a score of 8 or higher on the Demoralization Scale-II [27].

#### 3.3.2 Exclusion Criteria

- 1. Life expectancy <6 months (determined by the patient's non-study PMD)
- 2. Poor functional status (Palliative Performance Scale-v2 <60%).
- 3. Cognitive impairment (Montreal Cognitive Assessment ≤25)¹ or diagnosis of a neurodegenerative disorder.

Phase I – Study drug(s)


<sup>&</sup>lt;sup>1</sup> See reference 142. Milanini, B., et al., *The Montreal Cognitive Assessment (MoCA) to screen for cognitive impairment in HIV over age 60.* Journal of acquired immune deficiency syndromes (1999), 2014. **67**(1): p. 67.

Version date: 03 April 2018 Protocol CHR#15-17825

- 4. The regular use of psychotropic medications within 2 weeks of study participation, including antidepressants (such as serotonin-reuptake inhibitors, tricyclic antidepressants and monoamine oxidase inhibitors), anxiolytics, stimulants, antipsychotics, anti-epileptics, cannabis products and non-topical corticosteroids. Low dose (less than or equal to 50mg) TCAs prescribed for neuropathic pain are not considered psychotropic. Participants are prohibited from using these medications during the study, but do not need to demonstrate a period of psychiatric stability for 2 weeks prior to enrollment. Patients will be asked to refrain from consuming prescription analgesics or alcohol the day before, of, and after psilocybin sessions.
- 5. History of a psychotic disorder or a bipolar disorder (determined by SCID-5).
- 6. Family history of psychotic disorder or bipolar disorder (first or second degree relative).
- 7. Current, severe Major Depressive Episode (These individuals will be referred to standard-of-care treatment in the community).
- 8. History of active suicidal ideation with intent in the last 6 months (Suicidal ideation score >3and Reason for ideation >1 on C-SSRS); or a history of suicide attempt in the last 5 years with Actual lethality/Medical damage >0 or Potential lethality >0 (on C-SSRS).
- 9. Narcissistic personality disorder, moderate-to-severe (determined by SCID-5-PD).
- 10. History of Hallucinogen Use Disorder (*Moderate or Severe*) or Hallucinogen Persisting Perception Disorder (determined by SCID-5).
- 11. History of a seizure disorder.
- 12. CNS metastases or symptomatic CNS infection.
- 13. Clinically significant cardiovascular disease (CAD, CHF, arrhythmia); baseline QTc>450msec; uncontrolled hypertension (SBP>139mmHG or DBP>89mmHG if over 65 years old) or tachycardia (average HR>90bpm if over 65 years old) averaged over at least two measurements.
- 14. Supplemental oxygen requirement.
- 15. Insulin-dependent diabetes mellitus or poorly controlled non-insulin dependent diabetes mellitus (e.g., history of an episode of hypoglycemia or hospitalization for hyperglycemia on the current regimen).
- 16. Inadequate hepatic function (Total bilirubin > normal institutional limits, OR AST >3 upper institutional upper limit of normal, OR AST >3 upper institutional upper limit of normal), as determined by most recent laboratory tests.
- 17. Inadequate renal function as determined by eGFR < 30 mL/min/1.73 m2 (based on the MDRD equation) or CrCl < 30 mL/min (based on the C-G equation).
- 18. Concomitant dosing of psilocybin with known UGT1A10 and UGT1A9 inhibitors (e.g., diclofenac and probenecid) will be avoided. There is *no* exclusion criterion based on the use of medications or substances that are inhibitors or inducers of CYP450 enzymes.
- 19. The use of efavirenz (a.k.a, Sustiva or Atripla).
- 20. If deemed by clinical judgment of the study investigators to be unsafe for undergoing the intervention and/or inappropriate for participating in a therapy group.

### 3.4 Duration of Therapy

In the absence of treatment delays due to adverse events, treatment may continue for 8 weeks or until:

- Inter-current illness that prevents further administration of treatment
- Unacceptable adverse event(s)

<sup>1</sup> Individuals taking antidepressants, anxiolytics and stimulants will be presented with the option of tapering off, and remaining off, of their medication for the duration of the study, if their prescribing physician agrees with this course of treatment.

Phase I – Study drug(s) 

- Patients decides to withdraw from the study
- Significant patient non-compliance with protocol
- General or specific changes in the patients' condition render the patient unacceptable for further treatment in the judgment of the investigator.

### 3.5 Duration of Follow Up

Patients will be followed for 3 months after completion of treatment or removal from study, or until death, whichever occurs first. Patients removed from study for unacceptable treatment related adverse event(s) will be followed until resolution or stabilization of all treatment related adverse events.

#### 3.6 Randomization Procedures

Patients will not be randomized; this is an open-label pilot trial with one treatment arm.

### 3.7 Study Timeline

### 3.7.1 Primary Completion

The study will reach primary completion 36 months from the time the study opens to accrual.

### 3.7.2 Study Completion

The study will reach study completion 48 months from the time the study opens to accrual.

Phase I – Study drug(s) 

### 4 Study Drugs

### 4.1 Description, Supply and Storage of Investigational Drugs

### 4.1.1 Investigational Drug: Psilocybin

Psilocybin is available as a powder that can be encapsulated for oral administration.

#### Classification

Psilocybin is an indoleamine psychedelic and is one of the "classic psychedelics." It has a chemical structure similar to that of the neurotransmitter serotonin.

#### Mechanism of Action

Psilocybin is an agonist of serotonin 5HT2A, 2C and 1A receptors [92, 101].

#### <u>Metabolism</u>

After ingestion, psilocybin is rapidly dephosphorylated to psilocin, which is metabolized via oxidation and glucuronidation in the small intestine and the liver, and subsequently excreted renally [91, 93, 94].

#### Contraindications

Current safety standards for experimental psilocybin administration [24, 143] include providing a comfortable environment, the presence of supportive and non-directive therapists or research staff, and strict exclusion criteria. Beyond this basic principle, psilocybin should generally not be administered to individuals with a personal or family history of psychosis or bipolar disease, or individuals who are acutely suicidal. It should also not be administered to individuals with severe cardiovascular disease or CNS disease (metastases, a seizure disorder, or traumatic brain injury). Co-administration with medications associated with the serotonin syndrome [144] should be avoided.

#### Availability

Psilocybin is a Schedule I compound, and so requires a DEA Schedule I license to handle. For the purposes of this study, psilocybin is available from the laboratory of Dr. Roland Griffiths at Johns Hopkins University (IND#133202).

#### Storage and handling

Psilocybin is stored at 15-30°C. Each subject's dose will be, to the nearest milligram, as close as possible to that indicated by their actual bodyweight (e.g., 0.30mg/kg or 0.36mg/kg), with a maximum dose not to exceed that calculated for a BMI of 35 at that participant's height. The psilocybin will be provided to UCSF in powder form, and the UCSF Investigational Drug Service of the UCSF Department of Pharmacy Services will encapsulate the drug. The study drug will be stored in a secure vault in the Investigational Drug Service in the Inpatient Pharmacy in Moffitt-Long Hospital (505 Parnassus Ave, San Francisco).

#### Side Effects

Psilocybin is known to be physiologically safe at the doses proposed for this study, and is not addictive [92, 102]. Safe administration is dependent on using a supportive and structured administration protocol [24]. Psilocybin is known to possibly cause the following transient side effects: Anxiety, thought disorder, nausea, emesis, increase or decrease in heart rate, increase or decrease in blood pressure, and headache [18, 24, 91, 95, 145, 146]. Anxiety and thought disorder reactions appear to be dose-dependent, with higher doses associated with greater frequency of temporary anxiety and thought disorder reactions [138].

Phase I – Study drug(s) 

#### Version date: 03 April 2018

# <u>Clinical Safety Data</u> Psilocybin, in the form of psilocybe mushrooms, has been consumed by humans for ritual and healing purposes for at least hundreds of years [147]. The most extensive review of mid-

Century reports of the safety of the controlled, clinical uses of psychedelics, including psilocybin, found an overall low incidence of adverse events [103]. After clinical research with psilocybin in North America stopped in the 1970s, psilocybin continued to be used legally as a psychotherapy adjunct in Germany and Switzerland in the 1980s and 90s, but no comprehensive safety data are available from this period [104, 148].

Since the 1990s, hundreds of doses of psilocybin have been administered to humans in clinical trials and research laboratories across North America and Europe. Gouzoulis-Mayfrank et al found negligible acute effects on vital signs (heart rate, blood pressure, temperature) and neuroendocrine levels (cortisol, prolactin, growth hormone), but did find significant transient mental status changes in eight healthy volunteers administered a moderate dose (0.2mg/kg, with total dose <15mg) of oral psilocybin [149]. A review of results from the Vollenweider laboratory in Zurich, Switzerland found that in 110 subjects administered 1-4 lowto-high doses of oral psilocybin there were no detectable persisting adverse effects, and all acute adverse reactions (e.g., dysphoria or anxiety) were controlled with interpersonal support alone, meaning no pharmacologic or other medical interventions were necessary [143]. Moreover, several subjects who did report acutely distressful experiences later claimed in longterm follow up that these experiences had been "enriching". [143] A subsequent review from that laboratory found that among 261 subjects who received low-to-high doses of oral psilocybin, both mystical-type experiences and acute anxious reactions were strongly positively correlated with drug dose [150]. Importantly, anxious reactions were also strongly correlated with the experimental setting (more anxiety was reported if the subject underwent a PET scan during the experiment), which argues in favor of the idea that the risk of adverse events can be mitigated by providing a comfortable and supportive setting for drug administration. This laboratory's recent findings from 50 subjects [151], and another 25 subjects [152] receiving a moderate oral dose of psilocybin (0.16mg/kg po or 0.215mg/kg po) reported no adverse events, and found improvement in mood. In contrast to the PET study above, another laboratory in London found no adverse events when they administered moderate dose iv psilocybin to 15 healthy subjects with prior psychedelic experience while undergoing brain fMRI; these subjects reported improved well-being on 2-week follow up [141].

Grob et al conducted the first modern study on the use of psilocybin in subjects with advancedstage cancer [18]. Subjects received a single moderate dose (0.2mg/kg) of oral psilocybin with pre- and post-drug supportive psychotherapy. This was well-tolerated with subjects showing only mild transient increases in blood pressure and heart rate compared to active placebo; no subjects experienced acute anxiety during the experience; and subjects spontaneously requested that a second dosing session be added to the protocol. Since the Grob et al. study, two larger double-blind RCTs of psilocybin-assisted psychotherapy in cancer patients with anxiety or depression, conducted at NYU and Johns Hopkins, were published; they both reported no adverse reactions (e.g., headache, anxiety or psychosis-like symptoms) lasting longer than 24 hours [19, 20]. Separately, the Johns Hopkins laboratory has reported zero persisting psychological problems among the 54 subjects to whom they had administered high dose (>25mg po) oral psilocybin to by 2008 [24]. By October 2016, the Johns Hopkins team has had no significant adverse events after administering psilocybin to approximately 270 subjects over 560 drug treatment sessions, and emergent medications have never been needed to maintain the safety of the subjects nor the study therapists (Griffiths, personal communication 2016).

Oral psilocybin has also been administered to other clinical populations in modern controlled clinical settings with good safety outcomes. Of 9 subjects with OCD who were administered low-

Phase I – Study drug(s)


to-high doses of oral psilocybin, the only adverse event reported was transient hypertension [110]. Of 15 nicotine-dependent smokers receiving moderate-to-high doses of oral psilocybin, adverse events included acute anxiety, mild transient increases in hypertension and heart rate, and mild headaches [108]. Of 10 subjects with alcohol dependence administered moderate-to-high doses of oral psilocybin, the only adverse event reported was mild transient hypertension [107]. A recent open-label pilot study of 12 subjects with treatment-resistant depression, each receiving a low oral dose (10mg) followed one week later by a high dose (25mg) found transient anxiety, thought disorder, nausea and headache, but no severe or unexpected adverse events when followed for up to 3 months after the high dose session [153]. Finally, recent epidemiological data argue for a positive correlation between lifetime classic psychoelelic use (including psilocybin) in the US population and reduced rates of past month psychological distress, past year suicidal ideation and past year suicidal attempt [154].

#### 4.2 Drug Accountability

Each UCSF campus investigator using Schedule I substances in research must obtain their own Schedule I registration with the DEA and is responsible for the ordering, security, accountability and disposition of all product ordered under their registration. Psilocybin will be obtained from the laboratory of Dr. Roland Griffiths at Johns Hopkins University, and the drug will be shipped to the Investigational Drug Service of the Department of Pharmaceutical Services at UCSF Medical Center (505 Parnasssus Ave, Room M39C, San Francisco, CA 94143; Phone 415.353.1798). The pharmacy has been used for the storage and preparation of Schedule I controlled substances for individual campus Schedule I registrants for many years.

**Storage:** Schedule I substances will be stored in one of two large combination lock safes located in the investigational drug storage room of the UCSF Inpatient Pharmacy. The investigational drug storage room is a limited access storage room located in the basement of Moffitt Hospital on the UCSF Parnassus Campus (505 Parnassus Avenue). The room bears a security lock, accessible to the investigational pharmacy staff. The combination of the safe is known only to the investigational drug pharmacy staff.

Upon receipt of a medication order from the investigator, the drug supply will be accessed by the investigational pharmacy staff. The ordered dose will be obtained, placed in appropriate pharmacy dispensing container and labeled for the research subject. The dose contained will be sealed with a tamper evident seal. Research staff will escort the patient to the Inpatient Pharmacy on the day of dosing. Drug will be dispensed directly to the research subject by the pharmacy staff after confirming patient identification and acquiring the patient's signature on the pharmacy's chain of custody documentation. The subject will then be escorted by study staff from the Inpatient Pharmacy through indoor hallways that connect the Moffitt Hospital (where the pharmacy is located) to the Langley Porter Psychiatric Institute (where the drug administration will take place).

**Dispensing:** Psilocybin was shipped from Dr. Roland Griffiths in powder form and will need to be allocated into gelcaps by the UCSF Investigational Drug Service. Subjects will be dispensed one gelcap with their dose based on weight, as measured prior to the drug treatment day by study staff. Psilocybin will be ingested by study subjects in the testing area (Room A-310) of the third floor annex of Langley Porter Psychiatric Institute.

**Records:** Record keeping will be in accordance with federal and state regulations for Schedule I controlled substances. Inventory will be taken at least every two years at end of the business day and maintained in a printed form.

Phase I – Study drug(s) 

Version date: 03 April 2018 Protocol CHR#15-17825

### 4.3 Drug Ordering

UCSF has obtained psilocybin directly from Dr. Roland Griffiths at Johns Hopkins University.

### 4.4 Packaging and Labeling of Study Drugs

Drugs will be packaged and labeled per UCSF institutional standards, adhering to applicable local and federal laws.

Phase I – Study drug(s) 

#### 5 Treatment Plan

### 5.1 Dosage and Administration

Treatment will be administered on an outpatient basis.

**Table 5.1 Regimen Description** 

| Study<br>Drug | Premedication / precautions | Dose | Route | Schedule |
|---|---|---|---|---|
| Psilocybin | Avoid all other psychotropic agents within 48hr of each dose | 0.3mg/kg<br>or<br>0.36mg/kg<br>(moderate-<br>to-high) | Oral | After 4<br>group<br>therapy<br>visits |

Psilocybin is not physiologically toxic at the doses being used in this study. No human data exists that suggest what a toxic dose of psilocybin might be, but experiments in animals suggest that the LD50 of psilocybin in humans may be in the range of grams [91], which is two orders of magnitude higher than the highest dose to be used in this study. Patients could have short-term (<24hr) challenging psychological reactions. Patients who have a serious adverse event consisting of a negative psychological reaction lasting >24hr will be followed by a study physician until the resolution of the event and, at the discretion of the PI, may be removed from the study. There is reason to believe that participating in the integration group therapy sessions after a negative psychological reaction may help in recovering from such an event, and so participants will not automatically be removed from the study merely for having a prolonged negative psychological reaction to the psilocybin session (See Section 7.3 for definitions of Adverse Event.)

#### 5.1.1 Other Modalities

Patients will participate in group therapy sessions following a modified manual of Brief Supportive-Expressive Group Therapy (SEGT) [76]. SEGT emphasizes therapeutic goals that include enhancing mutual support, openness and emotional expression, improved social and family support, and detoxifying death and dying. The weekly sessions will last 90 minutes and be conducted by 2 co-facilitators with experience leading psychotherapy groups.

### 5.2 Monitoring and Toxicity Management

Of the hundreds of subjects administered psilocybin in clinical or research settings over the last two decades, none have required emergent psychiatric medications or emergency department care [24, 143, 154]. Each subject receiving psilocybin will be evaluable for safety. The safety parameters include physical findings and spontaneous reports of adverse events reported to the investigator by subjects and primary caregivers. Each subject will be assessed periodically for the development of any toxicity as outlined in <a href="Section 6 Study Procedures and Observations">Section 6 Study Procedures and Observations</a>. Toxicity will be assessed according to the NIH Division of AIDS Table of Grading of Severity of Adult and Pediatric Adverse Events V2.0 (http://rsc.tech-

res.com/Document/safetyandpharmacovigilance/DAIDS\_AE\_Grading\_Table\_v2\_NOV2014.pdf)

Phase I – Study drug(s) 

. We will monitor specifically for hypertension, hypotension, tachycardia, nausea, emesis, headache, anxiety, dysphoria, mania, suicidality and psychosis during drug sessions using the Adverse Event Medication Session Rating Form (see Appendix). Acute physical adverse events (e.g., nausea or hypertension) will trigger increased frequency of monitoring. Acute psychological adverse events will be managed by supportive reassurance and, if needed, medications such as lorazepam or olanzapine. Further management of physical or psychiatric adverse events will depend upon the judgment of the on-call study physician and may include, if necessary, transportation to the UCSF Parnassus Emergency Department, which is located immediately adjacent to the Langley Porter Psychiatric Institute.

Phase I – Study drug(s) 

#### 6 Study Procedures and Observations

See Appendix A for a timeline of all assessments

#### 6.1 Study Site

All in-person pre-treatment and treatment patient contact will occur at the Langley Porter Psychiatric Institute (LPPI) at 401 Parnassus Ave, San Francisco. LPPI is a psychiatric hospital within the UCSF Medical Center Parnassus Campus and is immediately adjacent to the UCSF Parnassus Emergency Department.

#### 6.2 Selection of Measures

Antiretroviral Medication Adherence Scale (AMAS)—A single item 11-point Likert scale (0%-100%) of ART medication adherence percentage over the past week. This scale was invented for this study.

Alcohol Use Disorders Identification Test (AUDIT) – A 10-item screening tool developed by the World Health Organization to assess alcohol consumption, drinking behaviors, and alcohol-related problems.

Center for Epidemiologic Studies Depression Scale-Revised (CES-D-R)—A 20-item validated 5-point Likert scale self-report scale for the detection of depression [155] that has been shown to be sensitive to change in symptoms in palliative care patients. [156].

Client Satisfaction Scale (CSS)—A 4-item 10-point Likert scale ("very dissatisfied" to "very satisfied") designed for this study assessing satisfaction with the intervention.

Clinical Global Impressions scale (CGI)—A widely-used 3-item clinician-administered assessment developed by the NIMH to assess change in patients in psychopharmacology trials[157].

Challenging Experiences Questionnaire (ChEQ)—A validated 26-item 6-point Likert scale of the extent to which subjects experienced challenging experiences during a psychedelic drug treatment session[158]. The scale has 7 factors: fear, grief, physical distress, insanity, isolation, death and paranoia.

Columbia Suicide Severity Rating Scale (C-SSRS)—A validated 17-item scale that assesses suicidal ideation and behavior (www.cssrs.columbia.edu) according to the Columbia Classification Algorithm for Suicide Assessment (C-CASA), which the FDA Division of Psychiatric Products requires be used in clinical trials it oversees.

Community Observer Rating Form (CORF)—A 13-item 10-point Likert scale developed by Griffiths et al to triangulate behavioral observations of individuals administered psilocybin [17].

Concomitant Therapeutics Checklist (CTC)—A checklist designed for this study to assess the following categories of mental health therapies used over the last week: Prescription medications, non-prescription medications, psychotherapy, mutual aid groups, self-help

Phase I – Study drug(s) 

techniques, integrative medicine modalities, other.

Credibility/Expectancy Questionnaire (CrEQ)—A 6-item self-report measure of cognitive and affective assessments of a mental health therapy with high internal consistency and good test-retest reliability [159] that we have adapted for psychological distress.

Demoralization Scale-II (DS-II)—An abbreviated, 16-item and 3-point version of the well-validated original 24-item Demoralization Scale [160], which is the most widely used self-report measure of demoralization in palliative care patients [29]. The DS-II has two subscales: Meaning and Purpose, and Distress and Coping Ability, and shows both good internal and external validity in palliative care patients [27, 161].

Drug Use Disorders Identification Test (DUDIT) – An 11-item screening tool developed as a parallel to the AUDIT to assess drug consumption, drug use behaviors, and drug-related problems.

Duke UNC Functional Social Support Questionnaire-5 (DUFSS-5)—A 5-item, 3-point Likert, self-report measure of perceived functional social support. The abbreviated 5-item scale has been validated in patients with severe medical illness (advanced cancer or AIDS) [162].

Experiences in Close Relationships scale—Modified 16 (ECR-M16)—A 16-item, 7-point Likert self-report measure of attachment security. The abbreviated 16-item version is reliable and has been validated in patients with severe medical illness (metastatic cancer)[163].

Group Questionnaire (GQ)—A validated self-report 30-item 7-point Likert questionnaire of therapeutic relationships in group therapy [130]. GQ has a three-factor model of group cohesion: Positive Bonding, Positive Working, Negative Relationships, all of which manifest in both member-member and member-leader relationships [164]. GQ was empirically-derived from measures in the AGPA CORE-R Battery [136] that assess therapeutic alliance and cohesion—the two factors known to best predict clinical outcomes of group psychotherapy trials [129].

Group Psychotherapy Intervention Rating Scale (GPIRS)—An empirically-derived observerrated 48-item instrument that assesses group therapist behaviors that help create and maintain group cohesion [165].

HIV and Abuse Related Shame Inventory (HARSI)—A validated 22-item 5-point Likert scale("Not at All" to "Very Much") (Neufeld et al 2012, AIDS Behavior, 16:1063-1074).

Hill Interaction Matrix (HIM)—The gold standard in group therapy process measures [166], the HIM is an observer-rated instrument that assesses group therapy sessions using a 4x4 matrix of style categories (conventional, assertive, speculative and confrontational) and content categories (general, group, personal, relationship). The HIM has been used since the 1960s and there exists an extensive database of normative data against which to compare outcomes [131].

International Personality Item Pool-Openness to Experience-20 (IPIP-OE-20)—A 20-item self-report measure that uses items in the public domain to evaluate a construct approximately equivalent to Openness, which is evaluated by the NEO-PI-R [167].

Inventory of Complicated Grief (ICG)—A well-validated 19-item 5-point Likert scale ("never" to "always") that is the gold standard self-report instrument for measuring complicated grief [168, 169].

McGill Quality of Life Questionnaire-Revised-Short (MQoL-RS)—A well-validated 15-item 11-point Likert scale that assess quality of life in palliative care patients by assessing the following

Phase I – Study drug(s) 

domains: Overall quality of life, Physical well-being, Psychological well-being, Social support and Existential well-being. We will only use 4 items, which are Parts A (Overall quality of life) and B (Physical symptoms).

Multidimensional Assessment of Interoceptive Awareness-Revised (MAIA-R)—A well-validated 32-item 6-point Likert scale of bodily and mental awareness that measures the following 8 domains: Noticing, Not-distracting, Not-worrying, Attention regulation, Emotional awareness, Self-regulation, Body listening and Trusting [170]. If this study, we will use the Emotional awareness (5-tiems), Self-regulation (4-items) and Trusting (3-items) subscales.

Mystical Experience Questionnaire-30 (MEQ-30)—A well-validated 30-item 6-point Likert scale ("none; not at all" to "extreme [more than any other time in my life]") self-report measure of mystical-type experiences [124], derived from the earlier work of Pahnke et al. [119].

Nature Relatedness Scale, Short-Form Version (NR-6)—A 6-item version of a well-validated 5-point Likert scale self-report measure of environmental connectedness (Nisbet, E. K., & Zelenski, J. M. (2013). The NR-6: a new brief measure of nature relatedness. Frontiers in Psychology, 4, 11. doi:10.3389/fpsyg.2013.00813)

Palliative Performance Scale version 2 (PPSv2)—A validated clinician-administered tool based on the Karnovsky Performance Scale but adapted for a palliative care population [113, 171].

Persisting Effects Questionnaire—Spirituality (PEQ-S)—An instrument developed by Griffiths et al for subjects who have been administered psilocybin to assess enduring changes in attitudes about life, attitudes about self, mood changes, relationships, behavioral changes, and spirituality [138]. The measure also includes 4 questions about the drug experience itself concerning personal meaningfulness, spiritual significance, how psychologically challenging it was, and personal psychological insights gained. We will only use the Spirituality subscale (59-item, 6 point Likert scale ["none; not at all" to "extreme"]), and the four questions about the psilocybin experience.

Post-traumatic Growth Inventory-Short Form (PTGI-SF)—A validated 10-item 6-point Likert scale meant to assess the following psychological factors in populations that have suffered a traumatic event or major crisis: quality of relationships with others, openness to new possibilities, personal strengths, spiritual change, and appreciation of life [172].

PTSD Checklist (PCL-5): A validated 20-item, 5-point Likert scale (from "Not at All" to "Extremely") to measure symptom criteria for PTSD from the DSM-5. [Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5)]

Quality of Life in Life Threatening Illness Family Caregiver version 2 (QoLLTI-Fv2)—A validated 17-item 11-point Likert scale (0-10) self-report measure that assesses seven domains of quality of life in caregivers for patients with life-threatening illness: state of carer, patient well-being, quality of care, outlook, environment, finances and relationships. This instrument was developed by the same laboratory that developed the McGill Quality of Life scale [173].

Schedule of Attitudes towards Hastened Death (SAHD)—A 20-item True/False self- report measure of the desire for hastened death validated in patients with HIV/AIDS and other palliative care conditions [174].

Social Connectedness Scale-Revised (SCS-R)—A well-validated 8-item 6-point Likert scale (negatively-worded items rated from "strongly agree" to "strongly disagree") self-report measure which has shown strong construct, convergent and discriminant validity as well as reliability ( $\alpha$  >

.92) for assessing the degree to which subjects feel connected to their social environment (Lee, R. M., & Robbins, S. B. (1995). Measuring Belongingness: The Social Connectedness and Social Assurance Scales. Journal of Counseling Psychology, 42(2), 232-241. doi:10.1037//0022-0167.42.2.232)

State-Trait Anxiety Inventory (STAI)—A 40-item 4-point Likert scale that is the gold standard in self-report measures for state and trait anxiety [175, 176].

Supportive-Expressive Group Therapy Topic Grid (SEGT-TG)—A measure developed by Spiegel and Spira for the original studies of SEGT[75]. Independent raters watch video of therapy sessions and document the number of minutes in which particular target discussion topics are handled in the session.

Structured Clinical Interview for DSM-5 (SCID-5)—The gold standard structured clinical interview for DSM-5 criteria for major psychopathology. We will use portions of the SCID to screen for lifetime Depressive, Psychotic, Bipolar and Hallucinogen-related disorders.

Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD)—A self-report questionnaire based on DSM-5 criteria for personality disorders. We will use this to screen for Cluster B personality disorders.

### 6.3 Qualitative Analyses

Qualitative analyses be grounded in Interpretive Phenomenological Analysis (IPA) [177]. Data for qualitative analysis will include transcripts from a convenience sample of group therapy sessions and psilocybin drug sessions, therapist process notes, patients' written accounts of their psilocybin experiences, verbal feedback elicited from patients throughout the study, transcripts from focus groups conducted after the study endpoint, and transcripts from 30-60 minute semi-structured interviews conducted with selected patients after the 6-month follow-up. IPA is widely used in studies of psychological interventions to better understand a patient's experience of their treatment, and is typically used to elicit convergent and divergent themes in studies with small sample sizes [177]. Two investigators with experience in qualitative analysis will at first independently code the same transcripts for prominent themes, followed by comparison of their codes until a consensus is reached on an appropriate coding scheme. A code book will be established which will be used to code further sources. Consensus will be reestablished on an iterative basis according to the criteria of the coders and the PI.

#### 6.4 Schedule of Procedures and Observations

The study-specific assessments are detailed in this section and outlined in Section 6 Schedule of Study Procedures and Assessments. Screening assessments will be performed on enrollment. Any results falling outside of the reference ranges may be repeated at the discretion of the investigator. All on-study visit procedures are allowed a window of  $\pm$  7 days unless otherwise noted. Treatment or visit delays for public holidays or weather conditions do not constitute a protocol violation.

A written, signed, informed consent form (ICF) and a Health Insurance Portability and Accountability Act (HIPAA) authorization must be obtained before any study-specific assessments are initiated. A copy of the signed ICF will be given to the subject and a copy will be filed in the medical record. The original will be kept on file with the study records.

### 6.4.1 Phone Screening

Phase I – Study drug(s)

Potential subjects will be screened over the phone to assure that they understand the time requirements of the study, they identify as a gay man, they are at least 50 years old, they were diagnosed with HIV prior to 1996, they report experiencing moderate-to-severe symptoms of demoralization on the DS-II and that they report complicated grief on the ICG, and that they do not meet any major exclusion criteria (e.g., history of psychosis or bipolar disorder; recent active suicidal ideation). A brief orientation to the study protocol, including psychoeducation on psilocybin, will be provided to patients who are not excluded. The patient will then be scheduled for an in-person screening and enrollment visit.

### 6.4.2 In-person Screening and Enrollment

Screening procedures and assessments to be completed on day of Enrollment (prior laboratory results from UCSF clinics may be considered instead of performing labs at enrollment if the results are less than 6 months old):

- Demographics questionnaire (Age, ethnicity/race, civil status, years of education, income)
- Vital signs; Physical examination; Complete medical and psychiatric history, including current medication list; Performance status (PPSv2); Mental Status Exam; Cognitive Status (Montreal Cognitive Assessment)
- Complete blood count (WBC, Hgb, Hct, Plt)
- Comprehensive metabolic panel (Na, K, Cl, CO2, BUN, Cr, Gluc, Tbili, Ast, Alt, AlkPhos, TProt, Alb)
- TSH, FT4
- Urinalysis
- Urine toxicology (must be completed on day of Enrollment)
- HIV viral load, CD4 count, CD8 count
- RPR or Treponemal Antibody
- Electrocardiogram (ECG)
- Selected screening portions of Structured Clinical Interview for DSM-5 Clinical Trials Version (SCID-5); sections on current Depressive disorders; lifetime Psychotic disorders, Bipolar disorders and Hallucinogen-related disorders), Structured Clinical Interview for DSM-5 Personality Disorders, self-report version (SCID-5-PD; section on Cluster B disorders)
- Columbia Suicide Severity Rating Scale (C-SSRS): Baseline/Screening (last 12 months)
- ART Medication Adherence Scale (AMAS), Centers for Epidemiologic Studies
  Depression Scale—Revised (CESD-R), Demoralization Scale—II (DS-II), Inventory of
  Complicated Grief (ICG), McGill Quality of Life Questionnaire-Revised-Short (MQoL-RS), PTSD Checklist-5 (PCL-5), Schedule of Attitudes towards Hastened Death
  (SAHD), State-Trait Anxiety Inventory (STAI).

Upon completing a successful in-person screening, subjects will also meet individually with one of the study therapists for 30 minutes to develop rapport and to discuss details about the subject's personal life, such as past and current relationships, family dynamics, and concerns about their disease. Finally, the subject will be placed on the waitlist until 6 subjects are available to start a group.

### 6.4.3 Baseline Assessments (Week 1)
Protocol CHR#15-17825

#### Version date: 03 April 2018

## 6.4.3.1 Baseline Subject Assessments

Baseline assessments will be filled out during an individual therapy session wherein the subject will meet one or both of the group therapists in the week prior to the first group therapy session. Separately, the subject's caregiver/important other will be invited to meet with study staff for a brief interview on their relationship with the subject [see Appendix C for interview guides]. The individual session for the study subject is meant to build trust and rapport with the group

therapists, to learn more about the subject's life history and struggles with his health, to elicit the subject's preferences and intentions for the treatment sessions, and to orient the subject further to the intervention protocol. If screening/enrollment measures were completed within 1 week of the baseline assessment, those measures will not need to be repeated.

 AMAS, AUDIT, CESD-R, CTC, DS-II, DUDIT, DUFSS-5, ECR-M16, ICG, IOS, IPIP-OE-20, MAIA-R, MQoL- RS, NR-6, PCL-5, PTGI-SF, SAHD, SCS-R, and STAI. A clinical rater will perform a CGI and C-SSRS(Interval) for each subject.

### 6.4.3.2 Baseline Caregiver/Important Other Assessments

CORF

#### 6.4.4 Treatment Period

#### 6.4.4.1 Group Therapy Sessions #1-4 (Weeks 2-3)

Patients will undergo four 90-minute group therapy preparatory sessions (2 per week) that will be audio and video recorded. Video footage of a random sampling of sessions will be analyzed with the HIM, SEGT-TG and the GPIRS. Patients will fill out the GQ after the sessions in Week 2 and 4. A clinical rater will administer the C- SSRS(Interval) to each subject at each weekly study visit.

# 6.4.4.2 Individual Drug Sessions (Weeks 4-5)

Patients will undergo individual drug sessions in which they are administered psilocybin 0.30mg/kg (or 0.36mg/kg) po, with a maximum dose not to exceed that calculated for a BMI of 35 at their height. The drug will be administered following the safety guidelines outlined by Johnson et al [24].

The day prior to the session, patients will be screened over the phone for contraindicated medications and reminded about procedures for the medication visit. Specifically, participants will be reminded that they cannot drive an automobile for the rest of the day after their medication visit, and they will be advised that if they will take the BART, they should not drive their car to the BART station.

On the day of the medication visit, patients will arrive at the Langley Porter Psychiatric Institute by 08:00 and be oriented to the drug session room, which will contain a couch for the patient to lie on and aesthetically pleasing décor. Before the medication session starts, participants will complete a urine drug screen and the CrEQ. Participants will then hand over their shoes, keys, wallet and phones to the study therapists for safe keeping; these will all be returned to the patient upon completion of the treatment session.

The entire session will be audio and video recorded for subsequent behavioral analysis and rating of therapist adherence to the therapy protocol. The patient will ingest the psilocybin capsules with 4 ounces of water and then be instructed to lie down on the couch wearing

Phase I – Study drug(s) 

Protocol CHR#15-17825

eyeshades and listening to a preselected music soundtrack via headphones. The subject will be instructed to focus their attention internally and to attempt to interact minimally with the two therapists who will be present in the room throughout the drug session, but will be as non-directive as possible in their interactions with the patient. In the event of a psychologically challenging experience such as significant anxiety or confusion, the therapists will provide verbal reassurance. Patients will have been instructed in the preparatory therapy session to notify the study therapists if during the treatment they feel anxiety or fear.

In the event of a psychiatric emergency, verbal de-escalation and physical and/or chemical restraint will be used to maintain the safety of the subject and the therapists, according to the clinical judgment of the on-call study physician. All possible efforts will be made to avoid using restraints of any kind. Subjects will not be allowed to leave the premises until the drug effects have worn off.

During the drug session, vital signs (heart rate and blood pressure) will be recorded at 10 minutes prior to drug ingestion, and then 30, 60, 90, 120, 180, 240, 300, and 360 minutes after drug ingestion.

In the event of a medical emergency, subjects will be evaluated by the on-call study physician who will be on-site for all drug administrations. At least one ACLS-certified study clinician will be on-site for all drug administrations. While expected to be rare, the most likely serious adverse event to occur would be a hypertensive crisis. If a subject's blood pressure becomes grossly elevated (SBP >180mmHg, DBP >110mmHG) or unsafe (BP elevations with associated symptoms such as chest pain or shortness of breath), blood pressure will be rechecked immediately in both arms and the on-call physician will be notified if s/he is not already in the treatment room. If the subject is clinically suspected of being in hypertensive emergency (with signs of end-organ damage), then the subject will be transported to the UCSF Emergency Department for further evaluation and treatment. The Emergency Department's door is less than a 1 minute walk from the Langley Porter Psychiatric Institute. If the patient if determined to be in hypertensive urgency (without clinical signs of end-organ damage), then blood pressure will be re-assessed every 5 minutes while the study physician continues to her/his evaluation for signs of clinical instability, and the study physician may attempt to calm the subject with verbal de-escalation or an anxiolytic (e.g. lorazepam) as transient hypertension is most likely to be due to a challenging psychological experience. If after 20 minutes the hypertensive urgency has not improved, the study physician will evaluate the need for transporting the subject to the Emergency Department for further evaluation and treatment. In the case of *acute chest pain*, the on-call study physician will have available sublingual nitroglycerin to administer to the subject and an electrocardiogram machine. A crash cart is located in the building, but the goal will be to transport a decompensating patient to the Emergency Department prior to the crash cart becoming imminently necessary. In the event of a suspected hypoglycemic episode in a subject with diabetes mellitus, a finger stick blood glucose will be checked on an as needed basis, and fruit or oral glucose tablets will be available.

As the drug effects begin to wear off at the 5-6 hour mark, the therapists will engage the patient in a therapeutic interview to explore the experience (see Appendix C for interview guide); this discussion will also be videotaped. A clinical rater will administer the C-SSRS(Interval). Only once patients are deemed to be free of the acute effects of the drug, and after at least 7 hours have passed since ingestion of the drug, will the participant be allowed to leave the premise in the company of a caregiver who has been instructed on how best to support the patient over the coming days.

The patient and caregiver will be given a study clinician's pager number in case of any clinical event off-site that needs further assessment. Patients must agree not to drive themselves home, nor to drive later that same day after they arrive home. Patients will be instructed to write a detailed account of their experience during the drug session at some point over the next week.

In the event that a participant did not arrange a friend/family member to accompany them home, the participant will be required to stay with the study clinicians longer, will be

Phase I – Study drug(s) 

encouraged to eat, and then the participant will be escorted to the curb by study staff and seen into a taxi/Lyft/Uber that will be instructed to take them home. The participant will also be instructed to call the study MD when they arrive home. All efforts will be made to avoid this situation. In the weeks prior to the medication session, participants will be regularly reminded to arrange for someone to accompany them home.

The following day patients will return to the study site to meet with a study therapist and engage in a therapeutic discussion of their experience for 90 minutes. Patients will complete the MEQ-30, ChEQ, STAI, SAHD, MQoL, and the C-SSRS(Interval) at this visit. Patients may again meet with study staff in person prior to the next group therapy session if they request this or if study clinicians deem it clinically warranted.

### 6.4.4.3 Group Therapy Sessions #5-10 (Weeks 6-8)

Patients will undergo six group therapy sessions each 90-minutes long. Video footage of a random sampling of sessions will be analyzed with the HIM, SEGT-TG, IGMIPS and the GPIRS. Prior to each session, patients will be screened for adverse events and evaluated with the CSSR-S. Prior to sessions 5, 7 and 9, participants will fill out the CTC. After sessions 6, 8 and 10, participants will fill out the GQ. At the end of session 5, participants will fill out these questionnaires: CESD-R, DS-II, ICG, PCL-5, HARSI. After sessions 7 and 10, participants will fill out the DS-II and ICG.

#### 6.4.5 Endpoint Assessments

## 6.4.5.1 Endpoint (Week 8) Study Measures for Subjects

Immediately after the last group therapy session (Week 8), patients will complete the AMAS, CESD-R, DS-II, DUFSS-5, ECR-M16, ICG, IOS, MQoL-RS, NR-6, PCL-5 SAHD, SCS-R, STAI, PTGI-SF, IPIP-OE-20, MAIA-R, HARSI, CTC, and CSS. A clinical rater will perform a MoCA and CGI for each subject.

# 6.4.5.2 Endpoint (Week 8) Study Measures for Caregivers/Important Others

Patients' primary caregivers/important others will complete the CORF and CSS.

# 6.4.6 Post-treatment/Follow Up Assessments

# 6.4.6.1 Focus Group (Week 10)

Two weeks after the last group therapy session, subjects and their caregivers/important others will be invited to participate in a focus group wherein they will be asked to give feedback regarding their experiences in the study. Effort will be made to get both responders and non-responders to attend the focus groups. A clinical rater will administer the C-SSRS(Interval) to each subject. Prior to the focus group each participant will fill out the DS-II and ICG. This will be video-recorded for subsequent qualitative analysis. See Appendix C for focus group guide.

# 6.4.6.2 3-Month Follow-up for Subjects

At 3 Months, patients will be mailed a packet with the following measures to be completed: AMAS, AUDIT, CESD-R, DS-II, DUDIT, DUFSS-5, ECR-M16, HARSI, ICG, MQoL-RS, NR-6, PCL-5, SAHD, SCS-R, STAI, PTGI-SF, IPIP-OE-20, MAIA-R, CTC, and the CSS. They will be called and encouraged to complete the packet.

Phase I – Study drug(s)


Version date: 03 April 2018 Protocol CHR#15-17825

## 6.4.6.3 3-Month Patients for Caregivers/Important Others

At 3 Months, primary caregivers/important others will be mailed a packet with the following measures: CORF and CSS. They will be called and encouraged to complete the packet.

#### 6.4.6.4 3-Month Qualitative Interviews

Between the Focus Group and the 3-month follow-up, subjects and caregivers/important others will be invited to participate in a semi-structured interview of their experience in the study. These interviews will be analyzed to detect potential mechanisms of the intervention as well as outcomes not addressed by the study measures. See Appendix C for interview guide.

## 6.5 Discontinuation of Therapy

The Investigator will withdraw a patient whenever continued participation is no longer in the patient's best interest. Reasons for withdrawing a patient include, but are not limited to, disease progression, the occurrence of an adverse event or a concurrent illness, a patient's request to end participation, a patient's non-compliance or simply significant uncertainty on the part of the Investigator that continued participation is prudent. There may also be administrative reasons to terminate participation, such as concern about a patient's compliance with the prescribed treatment regimen.

## 6.6 Dietary Restrictions

No dietary restrictions are included in the protocol.

#### 6.7 Prohibited Medications

Patients are prohibited from using medications from the following classes while enrolled in the study:

- Serotonin Reuptake Inhibitors (SSRIs and SNRIs)
- Tricyclic Antidepressants (TCAs)
- Monoamine Oxidase Inhibitors (MAOIs)
- Atypical antidepressants (e.g., mirtazapine, nefazodone)
- Antipsychotics/Neuroleptics (typical and atypical)
- Anti-epileptics or mood stabilizers (e.g., lithium, valproate)
- Stimulants (e.g., methylphenidate, modafinil)
- Efavirenz (Sustiva, in Atripla)
- Insulin
- Non-topical corticosteroids
- Herbal supplements intended to affect mood or anxiety.

#### Conditional medication restrictions

- Trazodone
  - Trazodone ≤50mg/24hr for insomnia is allowed, but not within 48hr of psilocybin session
- Benzodiazepines
  - o PRNs are allowed, but not within 48hr of psilocybin session
  - o "z-drugs" (e.g., zolpidem) are not allowed within 48hr of psilocybin session
- Non-benzodiazepine anxiolytics (e.g. gabapentin, buspar)
  - Gabapentin for neuropathic pain is allowed, but not within 48hr of psilocybin session

Individuals who at screening are excluded for taking contraindicated antidepressants, anxiolytics,

Phase I – Study drug(s) 

Version date: 03 April 2018 Protocol CHR#15-17825

stimulants or herbal supplements can be re-screened for the study if—under the guidance of their usual physician—they successfully taper off these medications and demonstrate a period of psychiatric stability lasting at least 2 weeks. One exception to the required 2 week period is for individuals taking low dose TCAs (≤50mg imipramine equivalent) for reasons other than depression or anxiety (e.g., peripheral neuropathy or insomnia). These individuals may, under the guidance of their usual physician, taper off these medications and then be enrolled in the study once they are no longer taking the TCA.

#### 6.8 Study Clinicians

Study clinicians (group therapists and treatment session guides) will be approved by a panel consisting of: Dr. Josh Woolley (PI), Dr. Alicia Danforth (UCLA psilocybin team, and lead clinical supervisor for UCSF the team), Dr. Brian Anderson (UCSF psilocybin team), and Robert Jesse (Johns Hopkins psilocybin team). Group therapists and treatment session guides will all be licensed clinicians (MD, RN, NP, MFT, LCSW, PhD, PsyD, Chaplain, etc) in the state of California; an exception will be made if the person is unlicensed but currently enrolled in a clinical training program and has had sufficient clinical exposure, according to the judgment of the above-mentioned panel. The selection of therapists/guides will give preference to those who have: 1) prior clinical experience working with the study population; 2) have demographic similarities to the study population (age, gender, sexual orientation); 3) prior experience conducting group therapy; 4) prior experience working with individuals under the influence of psychedelics either in research settings or harm-reduction settings (such as the Zendo Project); 5) have completed the CIIS certificate program in Psychedelic-assisted Psychotherapy and research; 6) must have completed CITI training and have been added to the study IRB.

Group therapist pairs will consist of one lead and one secondary therapist. The lead must have had significant experience as a group therapy leader; the secondary must have some experience as a group therapy leader. Group therapists will undergo at least 16 hours of training in Supportive-Expressive Group Therapy (SEGT) by studying SEGT training videos, the SEGT adherence rating scales that will be used in the study, and the 3 following SEGT manuals: the original manual for metastatic breast cancer patients [75], the manual for brief SEGT in newly diagnosed breast cancer patients [76], and the adaptation by Maldonado et al for patients with AIDS [78]. All group therapists will undergo at least one 'dry run' session of the SEGT method prior to starting a group.

Each subject will have 2 guides working with them in their drug treatment day (not necessarily one male and one female). At least one of the treatment session guides will be one of the subject's group therapy co-therapists. Treatment session guides will undergo instruction by Dr. Alicia Danforth and/or Dr. Anderson. Overall clinical supervision will be a responsibility shared by Dr. Josh Woolley (PI), Dr. Brian Anderson (lead medical supervisor) and Dr. Danforth (lead psychotherapy supervisor). Clinical consultation will be available from others involved in the study, such as Dr. Jim Dilley, Co-Investigator of this study and founder and of the UCSF Alliance Health Project, as well as Dr. Rob Daroff, a study clinician who is a staff psychiatrist at the SFVA with many years experiencing running psychotherapy groups for gay men in San Francisco.

Clinical supervision specifically related to psilocybin, and SEGT, will happen in the form of debriefing sessions after every study visit. Dr. Anderson will be an in-the-room observer of the group therapy sessions to take notes and later discuss with the group therapists their adherence to the SEGT method and its current adaptation to the psilocybin trial. Dr. Anderson and Dr. Danforth will review video of treatment sessions and discuss the technique observed with the

individual session guides on an as needed basis. Video segments of group therapy sessions and psilocybin treatment sessions will be used for discussion in a periodic supervision workshop to be held after the completion of each group therapy cohort and which all study clinicians will be highly encouraged to attend. The number of supervision sessions a study clinician is required to attend to maintain eligibility to work on the study will be up to the discretion of the clinical supervisors.

Phase I – Study drug(s)


## 7 Reporting and Documentation of Results

## 7.1 Evaluation of Safety and Feasibility

The assessment of safety and feasibility will be informed by surveillance of adverse events in all patients who enroll in the study. The study will use the NIH Division of AIDS Table of Grading of Severity of Adult and Pediatric Adverse Events V2.0 for reporting of adverse events. Analyses of feasibility and acceptability will also be informed by rates of patient recruitment and retention, therapist protocol adherence, self-report measures (CrEQ and CSS), and spontaneous feedback from subjects, caregivers/important others, and study therapists.

### 7.2 Evaluation of Efficacy

We will evaluate for trends in changes of group mean measures of demoralization, complicated grief, depression, anxiety, and other constructs mentioned above. These evaluations will consist of self-report measures (e.g., DS-II) and observations from caregivers/important others and clinical raters (e.g., CORF and CGI).

#### 7.3 Definitions of Adverse Events

#### 7.3.1 Adverse Event

An adverse event (also known as an adverse experience) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. More specifically, an adverse event (can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. An adverse event can arise from any use of the drug (e.g., off-label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.

#### 7.3.2 Adverse reaction

An adverse reaction is defined as any adverse event caused by the use of a drug. Adverse reactions are a subset of all suspected adverse reactions for which there is reason to conclude that the drug caused the event.

# 7.3.2.1 Suspected

A suspected adverse reaction is defined as any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, "reasonable possibility" indicates that there is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

# 7.3.2.2 Unexpected

An adverse event or suspected adverse reaction is considered *unexpected* if it is not listed in the investigator brochure or package insert(s), or is not listed at the specificity or severity that has been observed, or, if an investigator brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application.

"Unexpected," as used in this definition, also refers to adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs or

Phase I – Study drug(s) 

Version date: 03 April 2018 Protocol CHR#15-17825

as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

Adverse events that would be anticipated to occur as part of the disease process are considered *unexpected* for the purposes of reporting because they would not be listed in the investigator brochure.

#### **7.3.2.3 Serious**

An adverse event or suspected adverse reaction is considered *serious* if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death
- Life-threatening adverse event
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life function
- Congenital anomaly/birth defect

Important medical events that may not result in death, are life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

# 7.3.2.4 Life-threatening

An adverse event or suspected adverse reaction is considered *life-threatening* if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

# 7.4 Recording of an Adverse Event

All adverse events will be entered into UCSF REDCap, whether or not the event is believed to be associated with use of the study drug. Data about these events and their severity will be recorded using the NIH Division of AIDS Table of Grading of Severity of Adult and Pediatric Adverse Events V2.0.

The Investigator will assign attribution of the possible association of the event with use of the investigational drug, and this information will be entered into UCSF REDCap using the classification system listed below:

Phase I – Study drug(s) 

| Relationship | Attribution | Description |
|---|---|---|
| Unrelated to | Unrelated | The AE <i>is clearly NOT related</i> to the intervention |
| investigational drug/intervention | Unlikely | The AE <i>is doubtfully related</i> to the intervention |
| Deleted to | Possible | The AE <i>may be related</i> to the intervention |
| Related to investigational drug/intervention | Probable | The AE is likely related to the intervention |
| urug/intervention | Definite | The AE <i>is clearly related</i> to the intervention |

Signs or symptoms reported as adverse events will be graded and recorded by the Investigator. When specific adverse events are not listed in the above NIH DAIDS Table of Grading of Severity, they will be graded by the Investigator as *none*, *mild*, *moderate* or *severe* according to the following grades and definitions:

| Grade 0 | No AE (or within normal limits) |
|---|---|
| Grade 1 | Mild: Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated |
| Grade 2 | Moderate: Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated |
| Grade 3 | Severe: Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated |
| Grade 4 | Potentially life-threatening: Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death |
| Grade 5 | Death related to AE |

# 7.5 Follow-up of Adverse Events

All adverse events will be followed with appropriate medical management until resolved. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

# 7.6 Adverse Events Monitoring

All adverse events, whether or not unexpected, and whether or not considered to be associated with the use of the study drug, will be entered into UCSF REDCap, as noted above.

The Investigator will assess all adverse events and determine reportability requirements to the Data and Safety Monitor (DSM) and UCSF's Institutional Review Board, the Committee on Human Research (CHR); and, when the study is conducted under an Investigational New Drug Application (IND), to the Food and Drug Administration (FDA) if it meets the FDA reporting criteria.

In addition, all adverse events and suspected adverse reactions considered "serious," entered into UCSF REDCap will be reviewed and monitored by the Data and Safety Monitor on an

Phase I – Study drug(s) 

ongoing basis, discussed at DSM meetings which take place after each therapy group completes the 8-week intervention.

## 7.7 Expedited Reporting

#### Reporting to the Data and Safety Monitor

If a death occurs during the treatment phase of the study or within 30 days after the last administration of the study drug(s) and it is determined to be related either to the study drug(s) or to a study procedure, the Investigator or his/her designee must notify the DSM within 1 business day of knowledge of the event. The contact may be by phone or e-mail.

# Reporting to UCSF Committee on Human Research (Institutional Review Board)

The Principal Investigator must report events meeting the UCSF CHR definition of "Unanticipated Problem" (UP) within 10 business days of his/her awareness of the event.

## **Expedited Reporting to the Food and Drug Administration**

If the study is being conducted under an IND, the Sponsor-Investigator is responsible for determining whether or not the suspected adverse reaction meets the criteria for expedited reporting in accordance with Federal Regulations (21 CFR §312.32).

The Investigator must report in an IND safety report any suspected adverse reaction that is both serious and unexpected. The Sponsor-Investigator needs to ensure that the event meets all three definitions:

- Suspected adverse reaction (as defined in 7.3.2.1)
- Unexpected (as defined in 7.3.2.2)
- Serious (as defined in 7.2.3.3)

If the adverse event does not meet all three of the definitions, it should not be submitted as an expedited IND safety report.

The timeline for submitting an IND safety report to FDA is no later than **15 calendar days** after the Investigator determines that the suspected adverse reaction qualifies for reporting (21 CFR 312.32(c)(1)).

Any unexpected fatal or life-threatening suspected adverse reaction will be reported to FDA no later than **7 calendar days** after the Investigator's initial receipt of the information (21 CFR 312.32(c)(2)).

Any relevant additional information that pertains to a previously submitted IND safety report will be submitted to FDA as a Follow-up IND Safety Report without delay, as soon as the information is available (21 CFR 312.32(d)(2)).

# Reporting to Pharmaceutical Companies providing Study Drug

Serious adverse reactions will be reported to the Heffter Research Institute and the Usona Institute, which are consultants for this study.

Phase I – Study drug(s) 

#### 8 Statistical Considerations and Evaluation of Results

#### 8.1 Study Design

This open-label single-arm mixed-methods pilot study will use descriptive statistics and qualitative methods to evaluate safety and feasibility in terms of rates of adverse events, patient recruitment and retention, and feedback on the intervention's utility, content and duration. Given the small sample size of this study, small-to-medium effect sizes will likely be undetectable; and so descriptive statistics will be used to report changes in mean measures at baseline compared to the endpoint, and again at the 3-month follow-up. Exploratory ANOVAs will also be done to model changes in therapeutic process values (e.g., group cohesion) over time. Qualitative thematic analysis will also be used to evaluate verbal and written reports of patient and caregiver/important other experiences with the study in order to optimize implementation of the intervention in larger, future trials.

#### 8.1.1 Randomization

No randomization procedures will be used.

#### 8.1.2 Stratification Factors

No stratification procedures will be used.

#### 8.2 Determination of Sample Size and Accrual Rate

#### 8.2.1 Sample Size and Power Estimate

This pilot study of the safety and feasibility of psilocybin-assisted group therapy aims to enroll at least 18 subjects, and will have a maximum total sample size of 36. We estimate needing to enroll 18 subjects given attrition rates of up to 45% reported in trials of other group therapies for existential distress in palliative care patients [114]. For comparison, four different safety and feasibility pilot studies of psilocybin-assisted psychotherapy have been conducted over the last two decades, and have included 9, 10, 12 and 15 patients each [18, 107, 108, 110]. Four recently published feasibility pilot studies of meaning-focused group psychotherapies for palliative care patients have included 5, 11, 11, and 16 patients each [40, 178-180].

Group therapy studies should include at least 2 groups of at least 4-6 members [135], so we plan to have at least 8 subjects complete the intervention. We expect to be able to enroll at least 6 subjects every 6 months.

Because the proposed study is a pilot focused on investigating safety and feasibility, power calculations for efficacy measures are not indicated. Pilot studies are often used to estimate values that are then utilized in power calculations for full-scale trials. Indeed, we will estimate effect size (ES) and the intraclass correlation coefficient (ICC) [132] for the intervention based on our preliminary efficacy results. Group psychotherapy trials generally require large sample sizes to demonstrate statistical significance in change in efficacy measures given the likely interdependence of clinical outcomes when interventions are delivered in groups [132, 133]. Thus, future full-scale trials can utilize our estimates to derive adequate, and likely large, sample sizes.

Phase I – Study drug(s) 

#### 8.2.2 Replacement Policy

Study subjects who have been assigned to a group and drop out prior to the first group session can be replaced by a new subject who will be assigned to the same group. Subjects who drop out after the first group therapy session will not be replaced.

#### 8.2.3 Accrual estimates

The annual number of eligible patients is high given the size of the population of HIV-seropositive gay-identified men in the San Francisco Bay Area. In 2014, San Francisco reported 15,979 people living with HIV, 14,221 of whom were men who have sex with men, and 9,202 of whom are 50 and older [8]. If accrual falls short of expectations, advertising and recruitment efforts will be expanded.

#### 8.3 Interim Analyses and Stopping Rules

After the occurrence of one Adverse Event judged to be Severe and potentially related to the drug/intervention, enrollment will be stopped until a Safety Review has been completed and the appropriate protocol amendments implemented.

## 8.4 Analyses Plans

The study's biostatistician is Matthew Boden, Ph.D. Alongside the PI, Dr. Boden will be coresponsible for assuring that clinical data are correctly collected, stored and analyzed. He will work directly with the PI to assure that interpretations of these data are coherent and justified. Dr. Boden's professional interests are rooted in the research, evaluation and implementation of evidence-based treatments for complex and severe mental disorders. As a Health Science Specialist at the Center for Innovation to Implementation (Ci2i), Veterans Affairs (VA) Palo Alto Health Care System, Dr. Boden investigates the clinical effects and implementation of evidence-based psychosocial treatments for psychotic, anxiety, and substance use disorders. His research utilizes a variety of assessment (e.g., structured clinical interviews, biological assays) and statistical (e.g., linear mixed models, exploratory structural equation modeling) techniques. As a Senior Evaluator at the Program Evaluation and Resource Center (PERC), VA Office of Mental Health Operations (OMHO), Dr. Boden supports OMHO's nationwide program evaluation and quality improvement efforts.

# **8.4.1 Analysis Population**

All patients who enroll in the study will be included in analyses of safety and tolerability.

All patients who make any contact at all with the study (including those who are screened out over the phone) will be included in analyses of feasibility.

All patients who enroll in the trial will be included in analyses of efficacy. Repeated efficacy measures will be gathered and trended, regardless of missing data or protocol non-adherence.

All patients who participate in at least one group therapy session will be included in analyses of psychotherapeutic process.

# 8.5 Primary Analysis

Safety analyses will be performed for all patients who enroll in the study. The study will use the NIH Division of AIDS Table of Grading of Severity of Adult and Pediatric Adverse Events V2.0 to

Phase I – Study drug(s) 

classify adverse events. Descriptive statistics (percentages) will be reported for the incidence of any Adverse Events reported, including suicidality as measured by the C-SSRS. Median scores will also be calculated for total scores of the feasibility measures: CSS, CrEQ, and PEQ-S. The differences of mean pre- and post-treatment scores on the CORF will be calculated. Differences in individual pre- and post-treatment MoCA scores will be assessed for each individual. Therapist protocol adherence will be reported as a rate of discussion topic deviations from the protocol.

#### 8.5.1 Exploratory Analyses

Change in efficacy measures from pre-treatment to post-treatment to 3-month follow-up will be analyzed with descriptive statistics to represent trends in mean levels. Recognizing that the calculations will likely be underpowered, we will also perform ANOVAs of the secondary outcome measures. To assist in gauging the clinical relevance of these data relative to measurement error, and to overcome some of the limitations of the study's small sample size, Reliable Change Indices (RCI) will be calculated [181]. Data from efficacy measures will also be used to estimate effect sizes and intraclass correlation coefficients for use in larger, future studies.

Change in process measures (e.g., the HIM, QPIRS and GQ) over time will be analyzed with ANOVAs to assess the slopes of individual participants and of the whole sample.

Qualitative thematic analyses will be conducted according to the methods outlined in Section 6.3. Iterative inductive analyses will be performed with the aid of NVivo analytical software.

## 8.6 Study Results

Study results will be reported following the guidelines of the TREND Statement for reporting of results from non-randomized interventions [182]. The study biostatistician will oversee or review the interpretation of all the above analyses and descriptive statistics.

## 9 Study Management

## 9.1 Pre-study Documentation

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki as stated in 21 CFR §312.120(c)(4); consistent with GCP and all applicable regulatory requirements.

Before initiating this trial, the Investigator will have written and dated approval from the Institutional Review Board for the protocol, written informed consent form, subject recruitment materials, and any other written information to be provided to subjects before any protocol related procedures are performed on any subjects.

The clinical investigation will not begin until either FDA has determined that the study under the Investigational Drug Application (IND) is allowed to proceed or the Investigator has received a letter from FDA stating that the study is exempt from IND requirements.

The Investigator must comply with the applicable regulations in Title 21 of the Code of Federal Regulations (21 CFR §50, §54, and §312), GCP/ICH guidelines, and all applicable regulatory requirements. The IRB must comply with the regulations in 21 CFR §56 and applicable regulatory requirements.

## 9.2 Institutional Review Board Approval

The protocol, the proposed informed consent form, and all forms of participant information related to the study (e.g. advertisements used to recruit participants) will be reviewed and approved by the UCSF CHR (UCSF Institutional Review Board). The initial protocol and all protocol amendments must be approved by the IRB prior to implementation.

#### 9.3 Informed Consent

All participants must be provided a consent form describing the study with sufficient information for each participant to make an informed decision regarding their participation. Participants must sign the CHR-approved informed consent form prior to participation in any study specific procedure. The participant must receive a copy of the signed and dated consent document. The original signed copy of the consent document must be retained in the medical record or research file.

During enrollment, patients will be consented for participation in the study, including having the various aspects of their participation video-recorded. They will also sign a Release of Information for study staff to speak to the patients' primary caregivers and primary physicians. Primary caregivers/important others will also be consented during enrollment.

# 9.4 Changes in the Protocol

Once the protocol has been approved by the UCSF CHR, any changes to the protocol must be documented in the form of an amendment. The amendment must be signed by the Investigator and approved by the CHR prior to implementation.

If it becomes necessary to alter the protocol to eliminate an immediate hazard to patients, an amendment may be implemented prior to CHR approval. In this circumstance, however, the Investigator must then notify the CHR in writing within five (5) working days after implementation. The Study Chair and the UCSF study team will be responsible for updating any participating sites.

Phase I – Study drug(s) 

## 9.5 Handling and Documentation of Clinical Supplies

The UCSF Principal Investigator and each participating site will maintain complete records showing the receipt, dispensation, return, or other disposition of all investigational drugs. The date, quantity and batch or code number of the drug, and the identification of patients to whom study drug has been dispensed by patient number and initials will be included. The sponsor-investigator will maintain written records of any disposition of the study drug.

The Principal Investigator shall not make the investigational drug available to any individuals other than to qualified study patients. Furthermore, the Principal Investigator will not allow the investigational drug to be used in any manner other than that specified in this protocol.

## 9.6 Case Report Forms (CRFs)

The Principal Investigator and/or his/her designee, will prepare and maintain adequate and accurate participant case histories with observations and data pertinent to the study. Study specific Case Report Forms (CRFs) will document safety and treatment outcomes for safety monitoring and data analysis. All study data will be entered into UCSF REDCap via standardized CRFs in accordance with the CTMS study calendar, using single data entry with a secure access account. The Clinical Research Coordinator (CRC) will complete the CRFs as soon as possible upon completion of the study visit; the Investigator will review and approve the completed CRFs.

The information collected on CRFs shall be identical to that appearing in original source documents. Source documents will be found in the patient's medical records maintained by UCSF personnel. All source documentation should be kept in separate research folders for each patient.

In accordance with federal regulations, the Investigator is responsible for the accuracy and authenticity of all clinical and laboratory data entered onto CRFs. The PI will approve all completed CRFs to attest that the information contained on the CRFs is true and accurate.

All source documentation and CTMS data will be available for review/monitoring by the UCSF DSMC and regulatory agencies.

The Principal Investigator will be responsible for ensuring the accurate capture of study data. At study completion, when the CRFs have been declared to be complete and accurate, the database will be locked. Any changes to the data entered into the CRFs after that time can only be made by joint written agreement among the Study Chair, the Trial Statistician, and the Protocol Project Manager.

# 9.7 Oversight and Monitoring Plan

The DSM will routinely review all adverse events and suspected adverse reactions considered "serious". The DSM will audit study-related activities to ensure that the study is conducted in accordance with the protocol, local standard operating procedures, FDA regulations, and Good Clinical Practice (GCP). Significant results of the DSM audit will be communicated to the IRB and the appropriate regulatory authorities at the time of continuing review, or in an expedited fashion, as applicable. See Appendix for Data and Safety Monitoring Plan for additional information.

Phase I – Study drug(s) 

#### 9.8 Record Keeping and Record Retention

The Principal Investigator is required to maintain adequate records of the disposition of the drug, including dates, quantity, and use by subjects, as well as written records of the disposition of the drug when the study ends.

The Principal Investigator is required to prepare and maintain adequate and accurate case histories that record all observations and other data pertinent to the investigation on each individual administered the investigational drug or employed as a control in the investigation. Case histories include the case report forms and supporting data including, for example, signed and dated consent forms and medical records including, for example, progress notes of the physician, the individual's hospital chart(s), and the nurses' notes. The case history for each individual shall document that informed consent was obtained prior to participation in the study.

Study documentation includes all CRFs, data correction forms or queries, source documents, Sponsor-Investigator correspondence, monitoring logs/letters, and regulatory documents (e.g., protocol and amendments, CHR correspondence and approval, signed patient consent forms).

Source documents include all recordings of observations or notations of clinical activities and all reports and records necessary for the evaluation and reconstruction of the clinical research study.

In accordance with FDA regulations, the investigator shall retain records for a period of 2 years following the date a marketing application is approved for the drug for the indication for which it is being investigated; or, if no application is to be filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and FDA is notified.

#### References

- 1. High, HIV and Aging: State of Knowledge and Areas of Critical Need for Research. A Report of the NIH Office of AIDS Research by the HIV and Aging Working Group. J Acquired Immunodeficiency Syndrome, 2012. **60**(Suppl 1): p. S1-S18.
- 2. Brennan, M., et al., *A Needs Assessment of Older GMHC Clients Living with HIV*, ACRIA, Editor. n.d.
- 3. Applebaum, A.J., et al., *Future directions for interventions targeting PTSD in HIV-infected adults*. Journal of the Association of Nurses in AIDS Care, 2015. **26**(2): p. 127-138.
- 4. Parsons, J.T., et al., *Patterns of substance use among HIV-positive adults over 50: implications for treatment and medication adherence.* Drug and alcohol dependence, 2014. **139**: p. 33-40.
- 5. Ompad, D.C., et al., *Drug use among HIV+ adults aged 50 and older: findings from the GOLD II study.* AIDS care, 2016: p. 1-5.
- 6. Lovejoy, T.I., et al., Changes in sexual behavior of HIV-infected older adults enrolled in a clinical trial of standalone group psychotherapies targeting depression. AIDS and Behavior, 2015. **19**(1): p. 1-8.
- 7. Greene, M., et al., *Geriatric Syndromes in Older HIV-Infected Adults*. Journal of acquired immune deficiency syndromes (1999), 2015. **69**(2): p. 161-167.
- 8. San-Francisco-Department-of-Public-Health, HIV Epidemiology Annual Report. 2014.
- 9. Lee, V. and C.G. Loiselle, *The salience of existential concerns across the cancer control continuum.* Palliative and Supportive Care, 2012. **10**: p. 123–133.
- 10. Simms, V., I.J. Higginson, and R. Harding, *Integration of palliative care throughout HIV disease*. The Lancet infectious diseases, 2012. **12**(7): p. 571-575.
- 11. Yalom, I.D., Existential psychotherapy. 1980: Basic Books.
- 12. Kissane, D.W., *The relief of existential suffering*. Archives of internal medicine, 2012. **172**: p. 1501–1505.
- 13. Robinson, S., et al., A review of the construct of demoralization history, definitions, and future directions for palliative care. American Journal of Hospice and Palliative Medicine, 2016. **33**(1): p. 93-101.
- 14. Karpiak, S.E., R.A. Shippy, and M. Cantor, *Research on Older Adults with HIV*. 2006, AIDS Community Reserach Initiative of America: New York.
- 15. Neimeyer, R.A., *Meaning reconstruction & the experience of loss*. 2001: American Psychological Association.
- 16. Spitzer, M., et al., *Increased activation of indirect semantic associations under psilocybin.* Biological Psychiatry, 1996. **39**(12): p. 1055-1057.
- 17. Griffiths, R., et al., *Psilocybin can occasion mystical-type experiences having substantial and sustained personal meaning and spiritual significance*. Psychopharmacology, 2006. **187**: p. 268-83.
- 18. Grob, C.S., et al., *Pilot study of psilocybin treatment for anxiety in patients with advanced-stage cancer*. Archives of general psychiatry, 2011. **68**(1): p. 71-78.
- 19. Bossis, A.P., *Psilocybin-generated mystical experience research: Implications for alleviating existential distress associated with a cancer diagnosis. UCSF Osher Center.* October 2015: UCSF Osher Center.

- 20. American-College-Neuropsychopharmacology, *Active ingredient in magic mushrooms reduces anxiety, depression in cancer patients*, in *ScienceDaily*. 2015.
- 21. Jesse, R. and R. Griffiths, *Psilocybin Research at Johns Hopkins: A 2014 Report*, in *Seeking the Sacred with Psychoactive Substances*, J. Ellens, Editor. 2014, Praeger: Santa Barbara. p. 29-43.
- 22. Richards, W., et al., *LSD-assisted psychotherapy and the human encounter with death.* The Journal of Transpersonal Psychology, 1972. **4**: p. 121-150.
- 23. Soffer, J. and M.A. Cohen, *Psychotherapeutic Treatment of Psychiatric Disorders*, in *Handbook of AIDS Psychiatry*, M.A. Cohen, et al., Editors. 2010, Oxford University Press: New York. p. 201-217.
- 24. Johnson, M.W., W.A. Richards, and R.R. Griffiths, *Human hallucinogen research: guidelines for safety.* Journal of psychopharmacology, 2008. **22**: p. 603-620.
- 25. Classen, C.C. and D. Spiegel, *Supportive-Expressive Group Psychotherapy*, in *Handbook of Psychotherapy in Cancer Care*, M. Watson and D.W. Kissane, Editors. 2011, John Wiley & Sons, Ltd. p. 105-117.
- 26. Spiegel, D., Existential Psychotherapy for Patients With Advanced Cancer: Facing the Future and the Past. Journal of Clinical Oncology, 2015. **33**: p. 2713–2714.
- 27. Robinson, S., et al., *Refinement and revalidation of the Demoralization Scale: The DS-II-Internal Validity.* Cancer, 2016. **122**(14): p. 2251-2259.
- 28. Grob, C.S., A.P. Bossis, and R.R. Griffiths, *Use of the Classic Hallucinogen Psilocybin for Treatment of Existential Distress Associated with Cancer*, in *Psychological Aspects of Cancer*. 2013, Springer. p. 291-308.
- 29. Robinson, S., et al., A systematic review of the demoralization syndrome in individuals with progressive disease and cancer: a decade of research. Journal of pain and symptom management, 2015. **49**: p. 595–610.
- 30. Fang, C.-K., et al., A correlational study of suicidal ideation with psychological distress, depression, and demoralization in patients with cancer. Supportive Care in Cancer, 2014. **22**(12): p. 3165-3174.
- Puchalski, C., et al., *Improving the quality of spiritual care as a dimension of palliative care: the report of the Consensus Conference*. Journal of palliative medicine, 2009. **12**: p. 885–904.
- 32. Field, M.J., C.K. Cassel, and others, *Approaching Death:: Improving Care at the End of Life*. 1997: National Academies Press.
- 33. Frankl, V.E., *Man's search for meaning*. 1985: Simon and Schuster.
- 34. Yalom, I.D. and C. Greaves, *Group therapy with the terminally ill*. The American Journal of Psychiatry, 1977. **134**: p. 396-400.
- 35. Classen, C.C. and D. Spiegel, *Supportive-Expressive Group Psychotherapy*, in *Handbook of Psychotherapy in Cancer Care*. 2011, John Wiley & Sons, Ltd. p. 107-117.
- 36. Breitbart, W., et al., *Meaning-centered group psychotherapy: an effective intervention for improving psychological well-being in patients with advanced cancer.* Journal of Clinical Oncology: Official Journal of the American Society of Clinical Oncology, 2015. **33**: p. 749-754.
- 37. Henry, M., et al., *The Meaning-Making intervention (MMi) appears to increase meaning in life in advanced ovarian cancer: A randomized controlled pilot study.* Psycho-Oncology, 2010. **19**: p. 1340–1347.

- 38. Chochinov, H.M., et al., *Effect of dignity therapy on distress and end-of-life experience in terminally ill patients: a randomised controlled trial.* The lancet oncology, 2011. **12**: p. 753–762.
- 39. Kissane, D.W., et al., *Cognitive-existential group therapy for patients with primary breast cancer-techniques and themes.* Psycho-oncology, 1997. **6**: p. 25–33.
- 40. MacKinnon, C.J., et al., *A Pilot Study of Meaning-Based Group Counseling for Bereavement*. OMEGA Journal of Death and Dying, 2016. **72**(3): p. 210-233.
- 41. LeMay, K. and K.G. Wilson, *Treatment of existential distress in life threatening illness: a review of manualized interventions.* Clinical psychology review, 2008. **28**: p. 472–493.
- 42. Cassel, E.J., *The nature of suffering and the goals of medicine*. The New England journal of medicine, 1982. **306**: p. 639–645.
- 43. Hansen, N.B., et al., Longitudinal effects of coping on outcome in a randomized controlled trial of a group intervention for HIV-positive adults with AIDS-related bereavement. Death studies, 2006. **30**(7): p. 609-636.
- 44. Greene, M., et al., *Management of human immunodeficiency virus infection in advanced age.* Jama, 2013. **309**(13): p. 1397-1405.
- 45. Lennon, M.C., J.L. Martin, and L. Dean, *The influence of social support on AIDS-related grief reaction among gay men.* Social Science & Medicine, 1990. **31**(4): p. 477-484.
- 46. Martin, J.L. and L. Dean, *Effects of AIDS-related bereavement and HIV-related illness on psychological distress among gay men: A 7-year longitudinal study, 1985–1991.* Journal of consulting and clinical psychology, 1993. **61**(1): p. 94.
- 47. Cox, S., *The Legacy of the Past: Gay Men in Mid-Life and the Impact of HIV/AIDS*, M. Institute, Editor. 2006: New York.
- 48. Freiberg, M.S., et al., *HIV infection and the risk of acute myocardial infarction*. JAMA internal medicine, 2013. **173**(8): p. 614-622.
- 49. Silverberg, M.J., et al., *Cumulative incidence of cancer among persons with HIV in North America: a cohort study.* Annals of internal medicine, 2015. **163**(7): p. 507-518.
- 50. Heckman, T.G. and P.N. Halkitis, *Biopsychosocial aspects of HIV and aging*. Behavioral Medicine, 2014. **40**(3): p. 81-84.
- 751. Rosenfeld, B., et al., *Desire for hastened death among patients with advanced AIDS*. Psychosomatics, 2006. **47**(6): p. 504-512.
- 52. Julnes, P.S., et al., *The Association Between Post-traumatic Stress Disorder and Markers of Inflammation and Immune Activation in HIV-Infected Individuals With Controlled Viremia.* Psychosomatics, 2016. **57**(4): p. 423-430.
- 53. Skalski, L.M., et al., *Coping styles and illicit drug use in older adults with HIV/AIDS*. Psychology of Addictive Behaviors, 2013. **27**(4): p. 1050.
- 54. Halkitis, P.N., et al., *Psychosocial burdens negatively impact HIV antiretroviral adherence in gay, bisexual, and other men who have sex with men aged 50 and older.* AIDS care, 2014. **26**(11): p. 1426-1434.
- 55. Centers-for-Disease-Control-and-Prevention, HIV Surveillance Report, 2014. 2015.
- 56. Pence, B.W., *The impact of mental health and traumatic life experiences on antiretroviral treatment outcomes for people living with HIV/AIDS.* Journal of Antimicrobial Chemotherapy, 2009. **63**(4): p. 636-640.
- 57. Springer, S.A., A. Dushaj, and M.M. Azar, *The impact of DSM-IV mental disorders on adherence to combination antiretroviral therapy among adult persons living with HIV/AIDS: a systematic review.* AIDS and Behavior, 2012. **16**(8): p. 2119-2143.

- 58. Wagner, G.J., et al., *A closer look at depression and its relationship to HIV antiretroviral adherence*. Annals of Behavioral Medicine, 2011. **42**(3): p. 352-360.
- 59. Willie, T.C., et al., *Barriers to HIV medication adherence: examining distinct anxiety and depression symptoms among women living with hiv who experienced childhood sexual abuse.* Behavioral Medicine, 2016. **42**(2): p. 120-127.
- 60. Tsai, A.C., et al., *Directly observed antidepressant medication treatment and HIV outcomes among homeless and marginally housed HIV-positive adults: a randomized controlled trial.* American journal of public health, 2013. **103**(2): p. 308-315.
- 61. Tsai, A.C., et al., *Does effective depression treatment alone reduce secondary HIV transmission risk? Equivocal findings from a randomized controlled trial.* AIDS and Behavior, 2013. **17**(8): p. 2765-2772.
- 62. Negin, J., A. Rozea, and A.L. Martiniuk, *HIV behavioural interventions targeted towards older adults: a systematic review.* BMC public health, 2014. **14**(1): p. 1.
- 63. Justice, A.C., *HIV and aging: time for a new paradigm.* Current HIV/AIDS Reports, 2010. 7(2): p. 69-76.
- 64. Diverse-Elders-Coalition, *Eight policy recommendations for improving the health and wellness of older adults with HIV*. 2014.
- 65. Crisostomo, V., Personal communication (San Francisco AIDS Foundation). 2016.
- 66. Gokhale, K. *Drugs That Saved HIV Patients Now Threaten Them in Old Age*. 2016 6 July 2016; Available from: <a href="http://www.bloomberg.com/news/articles/2016-07-06/the-graying-face-of-hiv-spurs-race-to-simplify-therapies">http://www.bloomberg.com/news/articles/2016-07-06/the-graying-face-of-hiv-spurs-race-to-simplify-therapies</a>.
- 67. Bernstein, J., *What really killed Spencer Cox, AIDS activist?*, in *The New York Times*. 2013/02/22.
- 68. Bernstein, L., *The graying of HIV: 1 in 6 new U.S. cases are people older than 50*, in *The Washington Post*. 2016.
- 69. Brethauer, E. and T. Hussin, Last Men Standing. 2016.
- 70. Shumway, M., Personal communication. 2016.
- 71. Heckman, T.G., et al., *A randomized clinical trial of a coping improvement group intervention for HIV-infected older adults.* Journal of behavioral medicine, 2011. **34**(2): p. 102-111.
- 72. Sikkema, K.J., et al., *Outcomes from a randomized controlled trial of a group intervention for HIV positive men and women coping with AIDS-related loss and bereavement.* Death studies, 2004. **28**(3): p. 187-209.
- 73. Sikkema, K.J., et al., *A randomized controlled trial of a coping group intervention for adults with HIV who are AIDS bereaved: longitudinal effects on grief.* Health Psychology, 2006. **25**(5): p. 563.
- 74. Sikkema, K.J., et al., *Outcomes from a group intervention for coping with HIV/AIDS and childhood sexual abuse: reductions in traumatic stress.* AIDS and Behavior, 2007. **11**(1): p. 49-60.
- 75. Spiegel, D. and J. Spira, Supportive-Expressive Group Therapy: A Treatment Manual of Psychosocial Intervention for Women with Recurrent Breast Cancer. 1991: Stanford, CA.
- 76. Classen, C., et al., *Brief Supportive-Expressive Group Therapy for Women with Primary Breast Cancer*. 1993: Stanford.
- 77. Classen, C.C., et al., *Supportive–expressive group therapy for primary breast cancer patients: a randomized prospective multicenter trial.* Psycho-Oncology, 2008. **17**: p. 438–447.

- 78. Maldonado, J., et al., *Supportive-Expressive Group Therapy for People with HIV Infection: A Primer*. 1996: Stanford.
- 79. Heckman, T.G., Supportive-Expressive and Coping Group Teletherapies for HIV-Infected Older Adults: A Randomized Clinical Trial. AIDS Behavior, 2013. **19**(9): p. 3034-3044.
- 80. Kamen, C., et al., *The Impact of Stigma and Social Support on Development of Post-traumatic Growth Among Persons Living with HIV.* Journal of clinical psychology in medical settings, 2016: p. 1-9.
- 81. Willie, T.C., et al., *Anxiety and Depressive Symptoms Among People Living with HIV and Childhood Sexual Abuse: The Role of Shame and Posttraumatic Growth.* AIDS and Behavior, 2016: p. 1-12.
- 82. Sherr, L., et al., *HIV infection associated post-traumatic stress disorder and post-traumatic growth–a systematic review.* Psychology, health & medicine, 2011. **16**(5): p. 612-629.
- 83. Leserman, J., *Role of depression, stress, and trauma in HIV disease progression.* Psychosomatic Medicine, 2008. **70**(5): p. 539-545.
- 84. Sherman, A.C., et al., *Group interventions for patients with cancer and HIV disease: Part II. Effects on immune, endocrine, and disease outcomes at different phases of illness.*International journal of group psychotherapy, 2004. **54**(2): p. 203-233.
- 85. Ironson, G., H. Kremer, and A. Lucette, *Relationship Between Spiritual Coping and Survival in Patients with HIV.* Journal of general internal medicine, 2016: p. 1-9.
- 86. Ironson, G., et al., *Psychosocial and neurohormonal predictors of HIV disease* progression (CD4 cells and viral load): A 4 year prospective study. AIDS and Behavior, 2015. **19**(8): p. 1388-1397.
- 87. Löckenhoff, C.E., et al., *Five-factor model personality traits, spirituality/religiousness, and mental health among people living With HIV.* Journal of Personality, 2009. 77(5): p. 1411-1436.
- 88. Ironson, G.H., et al., *Personality and HIV disease progression: role of NEO-PI-R openness, extraversion, and profiles of engagement.* Psychosomatic Medicine, 2008. **70**(2): p. 245.
- 89. Moskowitz, J., et al., *Dispositional mindfulness in people with HIV: associations with psychological and physical health.* Personality and individual differences, 2015. **86**: p. 88-93.
- 90. Carod-Artal, F.J., *Hallucinogenic drugs in pre-Columbian Mesoamerican cultures*. Neurología (English Edition), 2015. **30**: p. 42–49.
- 91. Passie, T., et al., *The pharmacology of psilocybin*. Addiction biology, 2002. **7**(4): p. 357-364.
- 92. Nichols, D.E., *Psychedelics*. Pharmacological Reviews, 2016. **68**: p. 264-355.
- 93. Meyer, M.R. and H.H. Maurer, *Absorption, distribution, metabolism and excretion pharmacogenomics of drugs of abuse.* Pharmacogenomics, 2011. **12**: p. 215-233.
- 94. Hasler, F., et al., *Renal excretion profiles of psilocin following oral administration of psilocybin: a controlled study in man.* Journal of Pharmaceutical and Biomedical Analysis, 2002. **30**: p. 331-339.
- 95. Hasler, F., et al., *Acute psychological and physiological effects of psilocybin in healthy humans: a double-blind, placebo-controlled dose–effect study.* Psychopharmacology, 2004. **172**(2): p. 145-156.

- 96. Grinspoon, L. and J.B. Bakalar, *Psychedelic Drugs Reconsidered*. 1979, New York: Basic Books Inc.
- 97. Pahnke, W.N., *The psychedelic mystical experience in the human encounter with death.* Harvard Theological Review, 1969. **62**: p. 1–21.
- 98. Cohen, S., LSD and the anguish of dying, in Harper's Magazine. 1965. p. 69-78.
- 99. Barron, F., M. Jarvik, and S. Bunnell, *The Hallucinogenic Drugs*. Scientific American, 1964. **210**: p. 29-37.
- 100. Kast, E., *A Concept of Death*, in *Psychedelics: The Uses and Implications of Hallucinogenic Drugs*, B. Aaronson and H. Osmond, Editors. 1970, Anchor Books: Garden City. p. 366-380.
- 101. Nichols, D., *Hallucinogens*. Pharmacology & Therapeutics, 2004. **101**: p. 131-181.
- 102. MacLean, K.A., M.W. Johnson, and R.R. Griffiths, *Hallucinogens and Club Drugs*. The American Psychiatric Publishing Textbook of Substance Abuse Treatment, 2014: p. 209.
- 103. Strassman, R., *Adverse reactions to psychedelic drugs: A review of the literature*. The Journal of Nervous and Mental Disease, 1984. **127**: p. 577-595.
- 104. Passie, T., *Healing with entactogens*. 2012, Santa Cruz: Multidisciplinary Association for Psychedelic Studies.
- 105. Strassman, R.J., *Human psychopharmacology of N, N-dimethyltryptamine*. Behavioural brain research, 1995. **73**(1): p. 121-124.
- 106. MacLean, K.A., M.W. Johnson, and R.R. Griffiths, *Mystical experiences occasioned by the hallucinogen psilocybin lead to increases in the personality domain of openness.*Journal of Psychopharmacology, 2011. **25**(11): p. 1453-1461.
- 107. Bogenschutz, M.P., et al., *Psilocybin-assisted treatment for alcohol dependence: A proof-of-concept study.* Journal of Psychopharmacology, 2015. **29**: p. 289–299.
- 108. Johnson, M.W., et al., *Pilot study of the 5-HT2AR agonist psilocybin in the treatment of tobacco addiction.* Journal of Psychopharmacology, 2014: p. 0269881114548296.
- 109. Johnson, M.W., A. Garcia-Romeu, and R.R. Griffiths, *Long-term follow-up of psilocybin-facilitated smoking cessation*. The American Journal of Drug and Alcohol Abuse, 2016: p. 1-6.
- 110. Moreno, F.A., et al., *Safety, tolerability, and efficacy of psilocybin in 9 patients with obsessive-compulsive disorder*. Journal of Clinical Psychiatry, 2006. **67**(11): p. 1735-1740.
- 111. Griffiths, R., et al., *Mystical-type experiences occasioned by psilocybin mediate the attribution of personal meaning and spiritual significance 14 months later.* Journal of Psychopharmacology, 2008. **22**: p. 621-32.
- 112. Richards, W., Personal communication. 2016.
- Bakitas, M.A., et al., *Palliative care program effectiveness research: Developing rigor in sampling design, conduct, and reporting.* Journal of pain and symptom management, 2006. **31**: p. 270–284.
- 114. Applebaum, A.J., et al., Factors associated with attrition from a randomized controlled trial of meaning-centered group psychotherapy for patients with advanced cancer. Psycho-Oncology, 2012. 21: p. 1195-1204.
- 115. Breitbart, W., et al., *Meaning-Centered Group Psychotherapy: An Effective Intervention for Improving Psychological Well-Being in Patients With Advanced Cancer*. Journal of Clinical Oncology, 2015. **33**: p. 749–754.

- 116. Shilts, R., *And the band played on: People, politics, and the AIDS epidemic.* New York: St. Martins, 1987.
- 117. Leary, T., G.H. Litwin, and R. Metzner, *Reactions To Psilocybin Administered In A Supportive Environment.* The Journal of Nervous and Mental Disease, 1963. **137**: p. 561-573.
- 118. Blewett, D.B. and N. Chwelos, *Handbook for the Therapeutic Use of Lysergic Acid Diethylamide-25: Individual and Group Procedures*.

  <a href="https://www.erowid.org/psychoactives/guides/handbook\_lsd25.shtml">https://www.erowid.org/psychoactives/guides/handbook\_lsd25.shtml</a>. 1959.
- 119. Pahnke, W., et al., *The Experimental Use of Psychedelic (LSD) Psychotherapy*. JAMA, 1970. **212**: p. 1856-1863.
- 120. Preller, K.H., et al., *Effects of serotonin 2A/1A receptor stimulation on social exclusion processing*. Proceedings of the National Academy of Sciences, 2016. **113**(18): p. 5119-5124.
- 121. Dolder, P.C., et al., *Lsd acutely impairs fear recognition and enhances emotional empathy and sociality.* Neuropsychopharmacology, 2016. **41**(11): p. 2638-2646.
- 122. James, W., *The Varieties of Religious Experience*. 1902, New York: Modern Library.
- 123. Maslow, A., *Religions, Values and Peak Experiences*. 1964, Columbus: Ohio State University Press.
- 124. Barrett, F.S., M.W. Johnson, and R.R. Griffiths, *Validation of the revised mystical experiences questionnaire in experimental sessions with psilocybin*. Drug & Alcohol Dependence, 2015. **156**: p. e16.
- 125. Kurland, A.A., *LSD in the supportive care of the terminally ill cancer patient.* Journal of Psychoactive Drugs, 1985. **17**: p. 279-90.
- 126. Emerson, A., Personal communication. 2015.
- 127. Turton, S., D.J. Nutt, and R. Carhart-Harris, *A Qualitative Report on the Subjective Experience of Intravenous Psilocybin Administered in an fMRI Environment*. Current Drug Abuse Reviews, 2014. 7: p. 117-127.
- 128. Burlingame, G.M., A. Fuhriman, and J.E. Johnson, *Cohesion in group psychotherapy*. Psychotherapy: Theory, Research, Practice, Training, 2001. **38**: p. 373.
- 129. Burlingame, G.M., D.T. McClendon, and J. Alonso, *Cohesion in Group Therapy*, in *Psychotherapy Relationships that Work: Evidence-Based Responsiveness*, J.C. Norcross, Editor. 2011, Oxford University Press: Oxford.
- 130. Krogel, J., et al., *The Group Questionnaire: a clinical and empirically derived measure of group relationship.* Psychotherapy Research: Journal of the Society for Psychotherapy Research, 2013. **23**: p. 344-354.
- 131. Hill, W.F., *Hill interaction matrix*;: *A method of studying interaction in psychotherapy groups*. 3rd edition ed. 1965: Youth Study Center, University of Southern California.
- 132. Baldwin, S.A., D.M. Murray, and W.R. Shadish, *Empirically supported treatments or type I errors? Problems with the analysis of data from group-administered treatments.*Journal of consulting and clinical psychology, 2005. **73**: p. 924.
- 133. Fuhriman, A. and G.M. Burlingame, *Group psychotherapy: Research and practice*, in *Handbook of group psychotherapy: An empirical and clinical synthesis*, A. Fuhriman and G.M. Burlingame, Editors. 1994, John Wiley & Sons: New York.
- 134. Beck, A.P. and C.M. Lewis, *The Process of Group Psychotherapy: Systems for Analyzing Change*. 2000, Washington, D.C.: American Psychological Association.

- 135. American-Group-Psychotherapy-Association, *Practice Guidelines for Group Psychotherapy*. 2007.
- 136. Burlingame, G., et al., CORE Battery-Revised: An Assessment Tool Kit for Promoting Optimal Group Selection, Process and Outcome. 2006.
- 137. Kanas, N., *Group Therapy for Schizophrenic Patients*. 1996, Washington, D.C.: American Psychiatric Press Inc.
- 138. Griffiths, R., et al., *Psilocybin occasioned mystical-type experiences: immediate and persisting dose-related effects.* Psychopharmacology, 2011. **218**: p. 649–665.
- 139. Breitbart, W., et al., Meaning-centered group psychotherapy for patients with advanced cancer: A pilot randomized controlled trial. Psycho-Oncology, 2010. **19**: p. 21-28.
- 140. Shear, K., et al., *Treatment of complicated grief: a randomized controlled trial.* Jama, 2005. **293**(21): p. 2601-2608.
- 141. Carhart-Harris, R.L., et al., *Implications for psychedelic-assisted psychotherapy:* functional magnetic resonance imaging study with psilocybin. The British Journal of Psychiatry, 2012. **200**(3): p. 238-244.
- 142. Milanini, B., et al., *The Montreal Cognitive Assessment (MoCA) to screen for cognitive impairment in HIV over age 60.* Journal of acquired immune deficiency syndromes (1999), 2014. **67**(1): p. 67.
- 143. Studerus, E., et al., *Acute, subacute and long-term subjective effects of psilocybin in healthy humans: a pooled analysis of experimental studies.* Journal of Psychopharmacology, 2011. **25**: p. 1434–1452.
- 144. Boyer, E.W. and M. Shannon, *The Serotonin Syndrome*. New England Journal of Medicine, 2005. **352**: p. 1112-1120.
- Johnson, M.W., R.A. Sewell, and R.R. Griffiths, *Psilocybin dose-dependently causes delayed, transient headaches in healthy volunteers*. Drug and alcohol dependence, 2012. **123**: p. 132–140.
- 146. Carhart-Harris, R., et al., *The administration of psilocybin to healthy, hallucinogen-experienced volunteers in a mock-functional magnetic resonance imaging environment: a preliminary investigation of tolerability.* Journal of Psychopharmacology, 2011. **25**: p. 1562-1567.
- 147. Schultes, R.E., *Teonanacatl: The Narcotic Mushroom of the Aztecs*. American Anthropologist, 1940. **42**: p. 429–443.
- 148. Gasser, P. *Psycholytic Therapy with MDMA and LSD in Switzerland*. MAPS Bulletin, 1995. **5**, 3-7.
- 149. Gouzoulis-Mayfrank, E., et al., *Psychopathological, neuroendocrine and autonomic effects of 3, 4-methylenedioxyethylamphetamine (MDE), psilocybin and d-methamphetamine in healthy volunteers Results of an experimental double-blind placebocontrolled study.* Psychopharmacology, 1999. **142**(1): p. 41-50.
- 150. Studerus, E., et al., *Prediction of psilocybin response in healthy volunteers*. PLoS One, 2012. 7: p. e30800.
- 151. Kometer, M., et al., *Psilocybin-induced spiritual experiences and insightfulness are associated with synchronization of neuronal oscillations.* Psychopharmacology, 2015. **232**: p. 3663–3676.
- 152. Kraehenmann, R., et al., *Psilocybin-induced decrease in amygdala reactivity correlates with enhanced positive mood in healthy volunteers*. Biological psychiatry, 2015. **78**: p. 572–581.

- 153. Carhart-Harris, R.L., et al., *Psilocybin with psychological support for treatment-resistant depression: an open-label feasibility study.* The Lancet Psychiatry, 2016.
- 154. Hendricks, P.S., et al., Classic psychedelic use is associated with reduced psychological distress and suicidality in the United States adult population. Journal of Psychopharmacology, 2015. **29**: p. 280–288.
- 155. Eaton, W.W., et al., Center for Epidemiologic Studies Depression Scale: review and revision (CESD and CESD-R). 2004.
- Wakefield, C.E., et al., *Patient-reported depression measures in cancer: a meta-review.* The Lancet. Psychiatry, 2015. **2**: p. 635-647.
- 157. Guy, W., *ECDEU Assessment Manual for Psychopharmacology Revised.* 1976: Kensington, MD.
- 158. Barrett, F.S., et al., *The Challenging Experience Questionnaire: Characterization of challenging experiences with psilocybin mushrooms*. Journal of Psychopharmacology, 2016. **30**(12): p. 1279-1295.
- 159. Devilly, G.J. and T.D. Borkovec, *Psychometric properties of the credibility/expectancy questionnaire*. Journal of Behavior Therapy and Experimental Psychiatry, 2000. **31**: p. 73-86.
- 160. Kissane, D.W., et al., *The Demoralization Scale: a report of its development and preliminary validation.* Journal of palliative care, 2004. **20**: p. 269.
- 161. Robinson, S., et al., *Refinement and revalidation of the demoralization scale: The DS-II—external validity.* Cancer, 2016.
- 162. Saracino, R., et al., Measuring social support in patients with advanced medical illnesses: An analysis of the Duke-UNC Functional Social Support Questionnaire. Palliative & Supportive Care, 2015. 13: p. 1153-1163.
- 163. Lo, C., et al., Measuring attachment security in patients with advanced cancer: psychometric properties of a modified and brief Experiences in Close Relationships scale. Psycho-Oncology, 2009. **18**: p. 490-499.
- 164. Johnson, J., et al., *Group Climate, Cohesion, Alliance, and Empathy in Group Psychotherapy: Multilevel Structural Equation Models.* Journal of Counseling Psychology, 2005. **52**: p. 310-321.
- 165. Chapman, C.L., et al., *Rating group therapist interventions: The validation of the Group Psychotherapy Intervention Rating Scale.* Group Dynamics: Theory, Research, and Practice, 2010. **14**: p. 15.
- 166. Fuhriman, A. and G.M. Burlingame, *The Hill Interaction Matrix: Therapy Through Dialogue*, in *The Process of Group Psychotherapy: Systems for Analyzing Change*, A.P. Beck and C.M. Lewis, Editors. 2000, American Psychological Association: Washington, D.C. p. 135-174.
- 167. Goldberg, L., *The development of markers for the Big-Five factor structure*. Psychological Assessment, 1992. **4**: p. 26-42.
- 168. Shear, M.K., Complicated grief. N Engl J Med, 2015. 2015(372): p. 153-160.
- 169. Prigerson, H.G., et al., *Inventory of Complicated Grief: a scale to measure maladaptive symptoms of loss.* Psychiatry research, 1995. **59**(1): p. 65-79.
- 170. Mehling, W.E., et al., *The Multidimensional Assessment of Interoceptive Awareness* (MAIA). PloS One, 2012. 7: p. e48230.
- 171. Anderson, F., et al., *Palliative performance scale (PPS): a new tool.* Journal of palliative care, 1995. **12**: p. 5–11.

- 172. Cann, A., et al., A short form of the Posttraumatic Growth Inventory. Anxiety, Stress, & Coping, 2010. **23**(2): p. 127-137.
- 173. Cohen, R., et al., *QOLLTI-F: measuring family carer quality of life*. Palliative Medicine, 2006. **20**: p. 755-767.
- 174. Rosenfeld, B., et al., *Measuring desire for death among patients with HIV/AIDS: the schedule of attitudes toward hastened death.* American Journal of Psychiatry, 1999. **156**(1): p. 94-100.
- 175. Elwood, L.S., K. Wolitzky-Taylor, and B.O. Olatunji, *Measurement of anxious traits: a contemporary review and synthesis.* Anxiety, Stress, and Coping, 2012. **25**: p. 647-666.
- 176. Spielberger, C.D., State-Trait anxiety inventory. 2010: Wiley Online Library.
- 177. Brocki, J.M. and A.J. Wearden, *A critical evaluation of the use of interpretative phenomenological analysis (IPA) in health psychology.* Psychology & Health, 2006. **21**: p. 87-108.
- 178. Coward, D.D., Facilitation of self-transcendence in a breast cancer support group: II. Oncology Nursing Forum, 2003. **30**: p. 291-300.
- 179. van der Spek, N., et al., *Meaning-centered group psychotherapy in cancer survivors: a feasibility study.* Psycho-Oncology, 2014. **23**: p. 827-831.
- 180. Greenstein, M., *The house that's on fire: Meaning-centered psychotherapy pilot group for cancer patients.* American Journal of Psychotherapy, 2000. **54**: p. 501-511.
- 181. Jacobson, N.S., et al., *Methods for defining and determining the clinical significance of treatment effects: description, application, and alternatives.* Journal of Consulting and Clinical Psychology, 1999. **67**: p. 300-307.
- 182. Des Jarlais, D.C., et al., *Improving the reporting quality of nonrandomized evaluations of behavioral and public health interventions: the TREND statement.* American Journal of Public Health, 2004. **94**: p. 361-366.

| | | | WEEK 1 | WEEK 2 | WEEK 2 | WEEK 3 | WEEK 3 | WEEK 4-5 | WEEK 4-5 | WEEK 4-5 | WEEK 6 | WEEK 6 | WEEK 7 | WEEK 7 | WEEK 8 | WEEK 8 | FU:2Wee | kFU:3Mo | nth |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Phone Screen | Enrollment | Baseline + Meet Thrpsts | | | | | PSY-1day | | PSY+1day | | | G7 | G8 | G9 | G10 + Endpoir | | F/U | İ |
| Medical screening | | | | | | | | | | | - | | - | | - | | ,,,, | 1,75 | |
| History & Physical | | х | | | | | | | | | | | | | | | | | History & Physical |
| Labs | | х | | | | | | | | | | | | | | | | | Labs |
| ECG | | х | | | | | | | | | | | | | | | | | ECG |
| Urine drug screen | | х | | | | | | | x (pre) | | | | | | | | | | Urine drug screen |
| Phone Rx screen | | | | | | | | x | u/ | | | | | | | | | | Phone Rx screen |
| CLINICAL RATERS | | | | | | | | ~ | | | | | | | | | | | CLINICAL RATERS |
| MoCA | | x | | | | | | | | | | | | | | × | | | MoCA |
| PPSv2 | | x | | | | | | | | | | | | | | 1 | | | PPSv2 |
| SCID-5 | | х | | | | | | | | | | | | | | | | | SCID-5 |
| SCID-5-PD-B | | x | | | | | | | | | | | | | | | | | SCID-5-PD-B |
| ASI-Lite | | x | | | | | | | | | | | | | | | | | ASI-Lite |
| AE Screen | | - | x | x | х | x | x | x | x (during) | x | x | x | x | х | x | × | х | x | AE Screen |
| C-SSRS | | x | x | x | x | x | x | x | x(post) | x | x | x | x | x | x | × | x | x | C-SSRS |
| HIM | | | | x | x | x | x | | ( / | | x | x | | | x | x | | | HIM |
| GPIRS | | | | x | x | x | x | | | | x | x | | | x | × | | | GPIRS |
| SEGT-TG | | | | x | х | x | x | | | | x | x | | | x | × | | | SEGT-TG |
| STUDY THERAPISTS | | | | ~ | ^ | ^ | ^ | | | | ^ | ^ | | | | | | | STUDY THERAPISTS |
| BP/HR | | | | | | | | | x (during) | | | | | | | | | | BP/HR |
| CGI | | | x | | | | | | x (uu:g) | | | | | | | × | | | CGI |
| Process Notes | | | × | x | × | × | × | | × | × | × | x | | | × | × | | | Process Notes |
| SUBJECTS | | | ~ | _ | ~ | ^ | ^ | | | ~ | ^ | ^ | | | ^ | ^ | | | Measure |
| Demographics | | x | | | | | | | | | | | | | | | | | Demographics |
| GQ | | ^ | | | v | | v | | | | | v | | v | | v | | | GQ |
| СТС | | v | v | v | ^ | v | ^ | | x (pre) | | v | ^ | v | ^ | v | ^ | | v | СТС |
| AMAS | | v . | v | ^ | | ^ | | | х (ргс) | | ^ | | ^ | | ^ | v | | v . | AMAS |
| CESD-R | | v . | v | | | | v | | | | v | | | | | v | | v . | CESD-R |
| DS-II | v | ^<br>v | v | | | | v | | | | ^<br>v | | v | | | v | v | ^<br>v | DS-II |
| ICG | × | ^<br>v | v | | | | v | | | | ^<br>v | | v | | | v | v | ^<br>v | ICG |
| PCL-5 | | v | v | | | | v | | | | v | | ^ | | | v | ^ | v | PCL-5 |
| HARSI | | v . | v | | | | v | | | | v | | | | | v | | v . | HARSI |
| MQOL-RS | | v . | v | | | | v | | | v | ^ | | | | v | ^ | | v . | MQOL-RS |
| SAHD | | v . | v | | | | v | | | ^<br>v | | | | | v | | | v . | SAHD |
| STAI | | x | × | | | | × | | | × | | | | | × | | | x | STAI |
| ECR-M16 | | ^ | × | | | | ^ | | | | | | | | ^ | × | | x | ECR-M16 |
| AUDIT/DUDIT | | | X | | | | | | | | | | | | | 1 | | X | AUDIT/DUDIT |
| DUFSS-5 | | | × | | | | | | | | | | | | × | | | × | DUFSS-5 |
| IPIP-Openness-20 | | | × | | | | | | | | | | | | × | | | × | IPIP-Openness-20 |
| PTGI-SF | | Х | - | <b>†</b> | | | 1 | | | | l - | | 1 | 1 | x | <b>†</b> | | x | PTGI-SF |
| MAIA-R | | | x | <u> </u> | | | | | | | | | 1 | | x | 1 | | i i | MAIA-R |
| SCS-R | | | x | <b>†</b> | | | 1 | | | | l - | | 1 | 1 | х | <b>†</b> | | х | SCS-R |
| NR-6 | | | x | <b>†</b> | | | 1 | | | | l - | | 1 | 1 | x | <b>†</b> | | x | NR-6 |
| CrEQ | | | - | <b>†</b> | | | 1 | | x (pre) | | l - | | 1 | 1 | ľ. | <b>†</b> | | ř – | CrEQ |
| ChEQ | | | | <b>†</b> | | | 1 | | (5.0) | x | l - | | 1 | 1 | | <b>†</b> | | | ChEQ |
| MEQ-30 | | | | <b>†</b> | | | 1 | | | x | l - | | 1 | 1 | | <b>†</b> | | | MEQ-30 |
| CSS | | | | <b>†</b> | | | 1 | | | | l - | | 1 | 1 | | x | | x | CSS |
| Qualitative Interviev | v | х | | <b>I</b> | 1 | 1 | <b>†</b> | | | | <b> </b> | t | 1 | 1 | 1 | 1 | <b>†</b> | x | Qualitative Interview |
| Focus Group | | | | <b>†</b> | | | 1 | | | | l - | | 1 | 1 | | <b>†</b> | х | | Focus Group |
| CAREGIVER/IMPOR | TANT OTHER | | | | | | | | | | | | | | | | | | CAREGIVER/IMPORT OTHER |
| CORF | | | x | | | | | | | | | | | | | × | | х | CORF |
| CSS | | | - | <b>†</b> | | | 1 | | | | l - | 1 | 1 | 1 | | x | | x | CSS |
| Qualitative Interviev | v | | x | <b>I</b> | 1 | 1 | <b>†</b> | | | | <b> </b> | t | 1 | 1 | 1 | ľ. | <b>†</b> | x | Qualitative Interview |
| Focus Group | - | | | <del> </del> | <del> </del> | | <del> </del> | | | | <b> </b> | | <del> </del> | <del> </del> | 1 | <del> </del> | × | ř – | Focus Group |
| i ocus Group | | | l | l | l | I | l | | | | | l . | 1 | 1 | 1 | | ^ | 1 | i ocas oroup |